

### Statistical Analysis Plan

NCT Number: NCT05543174

Title: An Open-Label, Phase 3 Study to Evaluate the Efficacy and Safety of TAK-625 in

the Treatment of Subjects With Alagille Syndrome

Study Number: TAK-625-3001

Document Version and Date: Version 1.0 / 9-Sep-2025

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.



# STATISTICAL ANALYSIS PLAN for Final Analysis

Study Number: TAK-625-3001

Sable Terms of Use Study Title: An Open-Label, Phase 3 Study to Evaluate the Efficacy and Safety of TAK-625 in

Prepared by:

Based on:

Protocol Version: Amendment 2

Protocol Date: 08-Dec-2022

CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization broberty of Lay from Takeda.

### **REVISION HISTORY**

### **TABLE OF CONTENTS**

| 1.0 | OBJE | CTIVES, ENDPOINTS AND ESTIMANDS | 8 |
|---|---|---|---|
| 1.1 | | jectives | |
| | 1.1.1 | Primary Objective | 8 |
| | 1.1.2 | Primary Objective Secondary Objective(s) | <u>(e)</u> 8 |
| | 1.1.3 | Additional Objective(s) | <u>@</u> 8 |
| 1.2 | 2 En | dpoints | ,8 |
| | 1.2.1 | Additional Objective(s) dpoints Primary Endpoint(s) Secondary Endpoint(s) 2.2.1 Key Secondary Endpoints(s) | 8 |
| | 1.2.2 | Secondary Endpoint(s) | 8 |
| | 1.2 | 2.2.1 Key Secondary Endpoints(s) | 8 |
| | 1.2 | 2.2.2 Secondary Endpoint(s) | 8 |
| | | ¥ | |
| | 1.2.4 | Safety Endpoints | 10 |
| | 1.2.5 | Safety Endpoints Other Endpoints 2.5.1 PK Endpoint timand(s) Y DESIGN | 10 |
| | 1.2 | 2.5.1 PK Endpoint | 10 |
| 1.3 | B Est | timand(s) | 10 |
| 2.0 | STUD | Y DESIGN | 10 |
| 3.0 | STAT | ISTICAL HYPOTHESES AND DECISION RULES | 12 |
| 4.0 | SAMP | LE-SIZE DETERMINATION | 12 |
| 5.0 | ANAL | YSIS SETS | 12 |
| 5.1 | | Subjects Who Signed the Informed Consent Form | |
| 5.2 | 2 Al | Subjects Who Did Not Enter the Treatment Period | 12 |
| 5.3 | Sat | fety Analysis Set | 12 |
| 5.4 | | ention-to-treat set (ITT) | |
| 5.5 | | odified Intention-to-treat set (MITT) | |
| 5.6 | 6 Per | r-Protocol Analysis Set (PPS) | 13 |
| 6.0 | | STICAL ANALYSIS | |
| 6.1 | l X Ge | neral Considerations | 13 |
| 6.2 | An | alysis Approach | 15 |
| ,0 | 6.2.1 | Analysis Approach for Continuous Efficacy Endpoints | 15 |
| C | 6.2.2 | Analysis Approach for Binary Efficacy Endpoints | |
| | 6.2.3 | Analysis Approach for Time-to-Event Efficacy Endpoints | |
| 6.3 | B Dis | sposition of Subjects | 16 |
| | 6.3.1 | Study Information | 16 |
| | 632 | Disposition of Subjects | 16 |

| | 6.3.3 | Protocol Deviations and Analysis Sets | 17 |
|---|---|---|---|
| | 6.3. | 3.1 Significant Protocol Deviations | 17 |
| | 6.3. | 3.2 Analysis Sets | 18 |
| 6.4 | Con | comitant Medications | 18 |
| 6.5 | Exte | ent of Exposure and Compliance. | 19 |
| 6.6 | Effi | cacy Analysis | 19 |
| | G C | | 0.1 |
| 6.7 | | ety Analysis | 21 |
| | 6.7.1 | Adverse Events | |
| | 6.7. | 2 800 | |
| | 6.7. | | |
| | 6.7.2 | | |
| | 6.7. | 2.1 Laboratory Tests other than Urinalysis | 24 |
| | 6.7. | $\sim$ | 25 |
| | 6.7.3 | Vital Signs, Weight and Height | 26 |
| | 6.7.4 | ECGs. | |
| | 6.7.5 | Displays of Treatment-Emergent Adverse Events (Japanese) | |
| 6.8 | | rmacokinetic, Pharmacodynamic, and Biomarker Analyses | |
| | 6.8.1 | Pharmacokinetic Analysis | |
| | | ENCES | |
| | | GES TO PROTOCOL PLANNED ANALYSES | |
| | | DIX | |
| 9.1 | | nges From the Previous Version of the SAP | |
| 9.2 | ( ) | Handling Conventions | |
| | 9.2.1 | Definition of Study Days | |
| ζ^ | 9.2.2 | Definition of Study Visit Windows | |
| ,0 | 9.2. | 1 | |
| C) | 9.2. | 1 | |
| | 9.2. | | |
| | 9.2.3 | Partial Date Conventions | |
| 9.3 | | ivation of Endpoints | 33 |
| | 9.3.1 | Change from Week 18 to Week 22 of Primary and Secondary Efficacy | 2.2 |
| | | Endpoints | 33 |

| 9.3. | 2 ItchRO Average Scores | 33 |
|---|---|---|
| 9.3. | 5 Z-scores | -36 |
| 9.3 | 6 Lists of Laboratory Tests | 0 36 |
| 9.3. | 7 Table for AECI | 37 |
| 9.3. | 8 Significance Level and Confidence Coefficient. | 37 |
| 9.4 | Analysis Software | 37 |
| | 200 | |
| LIST OF I | 7 Table for AECI | |
| Table 9.1 | Visit Window of sBA | 29 |
| Table 9.2 | Visit Window of Liver Enzymes (ALT, ALP) and Bilirubins (Total and Direct) | |
| Table 9.3 | Visit Window of Vital Signs, Weight and Height, | 2) |
| | , CBC, Coagulation, Chemistry Panel, | |
| T 11 0 4 | Urinalysis, Serum Storage Samples Visit Window of ECGs | 30 |
| Table 9.4 | Visit Window of ECGs | 30 |
| Table 9.7 | Visit Window of Lipid Panel, Cholestasis Biomarkers (sBA subspecies, C4, FGF19, Autotaxin), Cipid Soluble Vitamins | |
| Table 9.8 | Visit Window of ItchRO Weekly Average Score | |
| | COL | |
| LIST OF I | IN-TEXT FIGURES | |
| Figure 2.1 | Sehematic Study Design | 12 |
| 1 | ede | |
| 101 | | |
| , ox | | |
| KX | | |
| Property of Lax | | |
| Richard | | |

### ABBREVIATIONS

ΑE adverse event

**AECI** adverse event of clinical interest

AFP alpha-fetoprotein **ALGS** Alagille syndrome ALP alkaline phosphatase **ALT** alanine aminotransferase **ANCOVA** analysis of covariance

aPTT activated partial thromboplastin time

AST aspartate aminotransferase 7αC4 7α-hydroxy-4-cholesten-3-one

BMI body mass index **BUN** blood urea nitrogen CBC complete blood count CI confidence interval

Electrocardiogram **ECG** 

fibroblast growth factor 19 FGF-19

gamma-glutamy/transferase **GGT** hepatocellular carcinoma **HCC** 

high density lipoprotein-cholesterol HDL-C

health-related quality of life HRQoL

ItchRO(Obs) ItchRO Observer ItchRO(Pt) ItchRO Patient

ITT intention-to-treat set

KM Kaplan-Meier

TDT-C low density lipoprotein-cholesterol

LIN lower limit of normal

last observation carried forward

Proper I c LS means least square means lipid soluble vitamin

**MCH** mean corpuscular hemoglobin

**MCHC** mean corpuscular hemoglobin concentration

Medical Dictionary for Regulatory Activities MedDRA

**MITT** modified intention-to-treat set **PEBD** partial external biliary diversion

PK pharmacokinetic

**PPS** per-protocol analysis set PRO patient-reported outcomes

PT preferred term 25th percentile Q1 Q3 75th percentile

QT interval corrected using Bazett's formula QTcB QT interval corrected using Fridericia's formula QTcF only and sul

QOL quality-of-life

retinol binding protein RBP SAE serious adverse event SAP statistical analysis plan

sBAserum bile acid

**SGOT** serum glutamic-oxaloacetic transaminase serum glutamic-pyruvic transaminase **SGPT** 

SOC system organ class

treatment-emergent adverse event **TEAE** 

triglycerides TG

WBC WHODrug do. total serum bilirubin **TSB** upper limit of normal white blood cell

World Health Organization Drug Dictionary

### 1.0

## 1.1

### 1.1.1

### 1.1.2

- To evaluate the PK of TAK-625 in subjects with ALGS.

  To evaluate the efficacy of TAK-625 on biochemical markers of cholestasts and liver disease in subjects with ALGS.

  Additional Objective(s)

  Applicable

  Endpoints

  Primary Endpoint

  2 change f

### 1.1.3

Not Applicable

### 1.2

### 1.2.1

The change from Week 18 to 22 of fasting sBA levels.

#### Secondary Endpoint(s) 1.2.2

#### Key Secondary Endpoints(s 1.2.2.1

- Change from baseline to Week 18:
  - $\Leftrightarrow$  Fasting sBA levels.
  - ♦ Pruritus as measured by ItchRO (Obs): weekly average severity (based on daily maximum of morning and evening severity scores).
  - Pruritus as measured by ItchRO (Obs): weekly average morning severity.
- Change from Week 18 to 22:
  - Pruritus as measured by ItchRO (Obs): weekly average severity (based on daily maximum of morning and evening severity scores).
  - Pruritus as measured by ItchRO (Obs): weekly average morning severity.

### Secondary Endpoint(s)

- Change from baseline to Week 18:
  - Pruritus as measured by Patient-reported Itch Reported Outcome (ItchRO [Pt]): weekly average severity (based on daily maximum of morning and evening severity scores).

- Change from Week 18 to 22:
- → Pruritus as measured by ItchRO (Pt): weekly average severity (based on daily maximum of morning and evening severity scores).

  → Pruritus as measured by ItchRO (Pt): weekly average morning

  → Liver enzymes (ALT and ALP) and L:1.



### 1.2.4 Safety Endpoints

- Incidence of AEs including SAEs, related to study drug, leading to study drug discontinuation, and AEs of clinical interest (AECIs).
  - *♦ AECIs include the following:*
  - *♦ LSV deficiency events.*
  - *♦ Liver parameter disruption.*
- Change from baseline in clinical laboratory values (hematology, chemistry, urinalysis, and others), physical examination findings (including body weight, height, and body mass index [BMI]), vital signs, and electrocardiogram (ECG) parameters.

### 1.2.5 Other Endpoints

### 1.2.5.1 PK Endpoint

- Plasma levels of TAK-625 at predose and approximately 4 hours after the morning dose at Week 12.
- Plasma levels of TAK-625 at predose (optional) and approximately 30 minutes after morning dose at Week 18 (or any visit up to Week 28).

### 1.3 Estimand(s)

Not Applicable.

### 2.0 STUDY DESIGN

This is a phase 3, multicenter, open-label, uncontrolled study to evaluate the efficacy and safety of TAK-625 in the treatment of Japanese subjects with ALGS.

### Study Population:

The study population is defined as "Japanese patients with ALGS who are 1 year of age or older".

Study Period (Screening, Treatment [Dose Escalation, Stable Dosing, and Follow-up Dosing], and Safety Follow-up Period):

This study consists of the screening period (up to 6 weeks prior to the study administration), 2-week dose escalation period (doses up to 400  $\mu$ g/kg/day, once a day [QD], as tolerated), 46-week stable dosing period, and follow-up dosing period (until TAK-625 is approved or available in Japan commercially, or if the subject withdraws from the study, or if the investigator determines the subject's discontinuation, or if the sponsor stops the program or development in this indication).

# 1. Screening Period (Up to 6 Weeks prior to the Study Administration):

In the screening period, for subjects who do not have documentation of mutation related to ALGS (JAGGED-1 or NOTCH2), genetic testing may be performed, if necessary. The electronic diary (eDiary) for assessing pruritus with the Itch Reported Outcome (ItchRO) instrument will be dispensed and subjects and caregivers will undergo training during the screening visit.

### 2. Dose Escalation Period (2 Weeks: Week 0 to 2):

In the 2-week dose escalation period, at the baseline visit (Week 0/Visit 2), subjects will be assessed to confirm continued study eligibility and undergo a physical examination including body weight, height, BMI, and vital signs, and have urine and blood samples taken for hematology, chemistry, fasting lipid panel, baseline levels of sBA, and other cholestasis biochemical markers. Compliance with ItchRO will be assessed. Study drug for Weeks 1 and 2 will be supplied at the baseline visit to eligible subjects. Subjects will receive the study drug, TAK-625, administered orally QD. The dose will be increased weekly over a 2-week period up to 400 μg/kg/day QD as follows: dose level 1, 200 μg/kg/day QD for 1 week; and dose level 2, 400 ug/kg/day OD for the remaining duration of the study. If an individual subject exhibits a treatment-emergent moderate or severe drug-related gastrointestinal (GI) toxicity with 400 ug/kg/day, study drug dose may be lowered to 200 ug/kg/day; later attempts to escalate the dose are permitted during the dose escalation period. This decision should be made in consultation with the medical monitor. If further dose escalations fail during the dose escalation period, the subject will remain on 200 μg/kg/day for the remainder of the study. The dose should be taken at least 30 minutes prior to the first meal of the day. It is recommended that the dose should be taken approximately at the same time each day for the duration of the treatment period. Subjects will return to the clinic at Week 3 and follow-up phone calls will be made at Weeks 1 and 2.

# 3. Stable Dosing Period (46 Weeks: Week 3 to 48):

After the dose escalation period, each subject will continue dosing with study drug at the Week 3 dose level, which is either 200 or 400 µg/kg/day, in the stable dosing period. Subjects will visit the study site at Weeks 6, 12, 18, 22, 28, 38, and 48, and undergo physical examinations. Subject contacts (phone calls) will be conducted as appropriate throughout the stable dosing period. Subjects and caregivers will continue twice daily completion of their ItchRO throughout the period.

# 4. Follow-up Dosing Period (after Week 48):

In the follow-up dosing period, each subject will continue dosing with study drug at the Week 48 dose level, which is either 200 or 400 µg/kg/day. The safety evaluation will be performed in all the subjects every 12 weeks from Week 48 visit until TAK-625 is approved or available in Japan commercially, or if the subject withdraws from the study, or if the investigator determines the subject's discontinuation, or if the sponsor stops the program or development in this indication. Bile acids and ItchRO will be measured to evaluate the long-term effectiveness of TAK-625. For subjects discontinuing early, safety follow-up will be conducted.

### 5. Safety Follow-up (after Final Visit/Early Termination [ET]):

Subjects/caregivers will have a final safety follow-up subject contact (phone call) 7 days after the final study visit or ET visit (except for screen failure).

A schematic of the study design is included as Figure 2.1.

Figure 2.1 **Schematic Study Design** 



#### 3.0 STATISTICAL HYPOTHESES AND DECISION RULES

Not Applicable.

### SAMPLE-SIZE DETERMINATION 4.0

ALGS is a rare disease. The targeted sample size is approximately 5 subjects based on enrollment feasibility of this population in Japan, rather than power calculation.

#### 5.0 **ANALYSIS SETS**

#### 5.1 All Subjects Who Signed the Informed Consent Form

All subjects who signed the informed consent form.

#### All Subjects Who Did Not Enter the Treatment Period 5.20

All subjects who did not enter the treatment period.

#### 5.3 Safety Analysis Set

All subjects who received at least one dose of study drug.

### 5.4 Intention-to-treat set (ITT)

All subjects who received at least one dose of study drug.

### **5.5** Modified Intention-to-treat set (MITT)

All subjects who received study drug through Week 18, and had a reduction from baseline in sBA levels of  $\geq$ 50% at the Week 12 or Week 18 measurement.

### 5.6 Per-Protocol Analysis Set (PPS)

All ITT subjects who did not have any of the following major protocol deviations and whose primary endpoint was evaluable.

- Subjects who did not meet inclusion criteria #3, 4, 6, or 10.
- Subjects who met exclusion criteria #2, 3, 4, 5, 6, 7, 14, 15, or 16.

### 6.0 STATISTICAL ANALYSIS

### **6.1** General Considerations

The following definitions and calculation formulas will be used.

- Treatment-emergent adverse event (TEAE): An adverse event whose date of onset occurs on or after the start of study drug.
- **Pretreatment event (PTE)**: Any untoward medical occurrence in a clinical investigation subject who has signed informed consent to participate in a study but prior to administration of study drug.
- **Descriptive statistics for endpoints**: Number of subjects, mean, standard deviation, standard error, maximum, minimum, and quartiles (Q1, median, and Q3).
- **Duration of exposure to study drug (days)**: {Date of last dose of study drug date of first dose of study drug + 1.
- **Duration of study after baseline (days)**: {Date of last visit/contact date of first dose of study drug} + 1.
- **Study drug compliance (%)**: Number of study drugs taken / duration of exposure to study drug\* 100 (rounded to 1 decimal place).
- Dose Level (μg/kg): Strength of study drug taken (mg) / (last available body weight (kg) prior to or on the day of study drug taken) \* 1000.
- Total Drug Exposure ( $\mu$ g/kg): Sum of {number of study drugs taken \* dose level received ( $\mu$ g/kg)}.
- **Average Daily Dose (μg/kg/day)**: Total Drug Exposure (μg/kg) / Duration of exposure to study drug (days).

- ItchRO (Obs/Pt) Daily Maximum of Morning and Evening Scores: Maximum of morning and evening severity scores for each day. The morning and evening severity scores of the same day should be used for the calculation. Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) itching.
- ItchRO (Obs/Pt) Daily Average of Morning and Evening Scores: Average of morning and evening severity scores for each day. The morning and evening severity scores of the same day should be used for the calculation. Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) itching.
- **Time to liver-associated events**: PEBD surgery, listing for liver transplantation, liver decompensation [hepatic encephalopathy, variceal bleeding, ascites, and spontaneous bacterial peritonitis] events, hepatocellular carcinoma (HCC), death, and other.
- Estimated Total Lipids (mg/dL): Cholesterol (mg/dL) + Triglycerides (mg/dL).
- Ratio of Alpha-tocopherol to Estimated Total Lipids (mg/g): 1000 \* Alpha-tocopherol (mg/dL) / Estimated Total Lipids (mg/dL). For Alpha-tocopherol concentrations reported as below the minimum quantitation limit, half of the minimum quantitation limit is used in the calculation.
- Corrected Sodium (mEq/L): sodium (mEq/L) + (0.002 \* Triglycerides (mg/dL)).

- Subject Type: [all subjects including ones under 1 year old (overall), 1 year or older].
- Time Since Original Diagnosis of ALGS (months): (date of first dose date of original diagnosis of ALGS + 1) / 30.44.
- **Significant Protocol Deviation**: Deviation defined in the PDMP as "Important PD" whose Severity Classifications is "major" or "critical".

When reporting derived values or parameters, following presenting rules will be applied.

- For sBA, ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.
  - For measures of median and mean, use 3 decimal places.
  - For measures of standard deviation, standard error of the mean and CI, use 4 decimal places.
  - For measures of minimum and maximum values as well as observed value (for Listing), use 2 decimal places.

- >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
- For p-values use 3 decimal places.
- Presentation of p-values display p-values that would round to 0.000 as <0.001.
- Other than sBA, and ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.
  - For measures of median and mean, use 1 decimal place beyond those used for the measurement.
  - For measures of standard deviation, standard error of the mean and CI, use 2 decimal places beyond those used for the measurement.
  - For measures of minimum and maximum values, use the same number of decimal places as those used for the measurement.
  - >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
  - For p-values use 3 decimal places.
  - Presentation of p-values display p-values that would round to 0.000 as <0.001.
  - ➤ BMI should be rounded to 1 decimal place for reporting.
  - ➤ Derived questionnaire scores, and other similar efficacy parameters recorded as integers, should be rounded to 1 decimal place for reporting.
  - Averaged lab results (e.g. Diastolic/Systolic Blood Pressure and Pulse [when taken in triplicate]) should be rounded to 1 decimal place for reporting.

# 6.2 Analysis Approach

# 6.2.1 Analysis Approach for Continuous Efficacy Endpoints

For efficacy endpoints, all continuous endpoints in this trial will use the analysis method below unless stated otherwise in the section specific to an endpoint.

- Change from Week 18 to Week 22:
  - Descriptive statistics and two-sided 95% confidence interval of mean will be provided for observed values (Week 18 (LOCF) and Week 22) and changes from Week 18 (Week 22 Week 18 (LOCF)) by subject type. For endpoint with multiple visits, these will be provided by visit.
- Change from baseline to post-baseline:
  - ♦ Descriptive statistics and two-sided 95% confidence interval of mean will be provided for observed values (baseline and post-baseline visits) and changes from baseline (each post-

Analysis Approach for Binary Efficacy Endpoints

For efficacy endpoints, all binary endpoints in this trial will use the analysis method below unless stated otherwise in the section specific to an endpoint.

• Frequency distribution will be provided by visit. with a confidence interval by subject the section of the subject the section of the subject the section of by visit.

#### 6.2.3 Analysis Approach for Time-to-Event Efficacy Endpoints

For efficacy endpoints, all time-to-event endpoints in this study will use the analysis method below unless stated otherwise in the section specific to an endpoint.

The event-free survival rate and the two-sided 95% confidence intervals will be provided using the Kaplan-Meier method. The event-free survival rate will also be plotted. Time to event will be defined as the date of first dose of study drug to the event which comes fastest. For subjects without an event, time to event will be defined as the date of first dose of study drug to the censoring date, which is the date of the last study visit/contact.

#### **Disposition of Subjects** 6.3

#### 6.3.1 **Study Information**

Analysis Set: All Subjects Who Signed the Informed Consent Form

Date First Subject Signed Informed Consent Form Analysis Endpoint(s):

Date of Last Subject's Last Visit/Contact

MedDRA Dictionary Version

WHO Drug Dictionary Version

SAS Version Used for Creating the Datasets

Analytical Method(s): (1) Study Information

Study information shown in the analysis endpoints section will be

provided.

### **Disposition of Subjects**

Analysis Set: ITT

Analysis Endpoint(s): [Completed Study Drug, Prematurely Study Drug Completion

> Status Discontinued Study Drug

Reason for Discontinuation

of Study Drug

[AE, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Lack of Efficacy, Other]

Completion Status of All Planned Study Visits

[Completed Study, Prematurely

Discontinued Study]

Reason for Discontinuation

of Study

[AE, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Lack of Efficacy, Other]

Analytical Method(s):

(1) Disposition of Subjects

Frequency distributions will be provided by subject type. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the

denominator.

#### **Protocol Deviations and Analysis Sets** 6.3.3

6.3.3.1 Significant Protocol Deviations

Analysis Set:

ITT

Analysis Endpoint(s):

Significant Protocol Deviation [Informed Consent and Process. Inclusion Criteria, Exclusion Criteria, Concomitant Medication, Laboratory Assessment, Study Procedures (not safety and efficacy related), Safety, Visit Schedule, IP conditions, IP preparation, IP administration, Subject IP Compliance, Efficacy,

Subject Discontinuation,

Administrative, Patient Reported Outcomes, PK/PD, Other Criteria]

(1) Protocol Deviations

Analytical Method(s): (1) Frequency distribution will be provided for each deviation category by subject type. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be

6.3.3.2 Analysis Sets

ITT Analysis Set:

Analysis Endpoint(s):

[Categories are based on the definitions in Section 5.0] Handling of Subjects the applicable

**Analysis Sets** 

ITT [Included] **MITT** [Included] **PPS** [Included] Safety Analysis Set [Included]

(1) Subjects Excluded from Analysis Sets Analytical Method(s):

(2) Analysis Sets

Frequency distributions will be provided by subject type. For (1), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted

only once.

#### 6.4 **Concomitant Medications**

Analysis Set:

Medication History Analysis Endpoint(s):

Concomitant Medications

Proberty of Lakeda. For Analytical Method(s) (1) Concomitant Medications That Started Prior to and Were

Ongoing at Baseline as well as Those That Started After Baseline by Anatomical Therapeutic Chemical Level 2 and Preferred

Medication Name

Frequency distributions will be provided by subject type. WHO Drug dictionary will be used for coding. Summaries will be provided using anatomical therapeutic chemical level 2 and preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication names will be counted only once for that preferred medication names. For anatomical therapeutic chemical level 2, same manners in counting frequency.

#### 6.5 **Extent of Exposure and Compliance**

ITT Analysis Set:

Analysis Endpoint(s): Duration of Exposure to

Study Drug (days)

= 14, 15 <= - <= Max]

[Min<= - <80, 80 <= - <= 100, 100 <- <= Max] Study Drug Compliance (%)

Total Drug Exposure (µg/kg)

Average Daily Dose

(µg/kg/day)

(1) Study Drug Exposure, Compliance, Total Drug Exposure and Analytical Method(s):

Average Daily Dose

Frequency distributions for categorical endpoints and descriptive statistics for continuous endpoints will be provided by subject type.

#### 6.6 **Efficacy Analysis**







# 6.7 Safety Analysis

### **6.7.1** Adverse Events

6.7.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): TEAE
Categories: Relation
Interest

Categories: Relationship to Study Drug [Related, Not Related]

Intensity [Mild, Moderate, Severe]

The following summaries will be provided by subject type. Analytical Method(s):

- (1) Overview of Treatment-Emergent Adverse Events
  - 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 2) Relationship of Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
  - 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 4) Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
  - 5) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 6) Relationship of serious Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
  - 7) Serious Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
  - Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below.

# Number of subjects

- Property of Takedai. For nord Summaries for 2) and 6) A subject with occurrences of TEAE in both categories (i.e., Related and Not Related) will be counted once in the Related category.
  - Summary for 3) A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.
  - Summaries other than 2), 3), and 6) A subject with multiple occurrences of TEAE will be counted only once.

### Number of events

For each summary, the total number of events will be calculated.

CONFIDENTIAL

#### 6.7.1.2 Displays of Treatment-Emergent Adverse events

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): **TEAE** 

Categories: Intensity [Mild, Moderate, Severe]

> [1-14, 15-169, 170-336,Time of Onset (day)

The following summaries will be provided using frequence Analytical Method(s):

distribution by subject type.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- Organ Class

  Into Emergent Adverse Events by System

  Intensity of Treatment-Emergent Adverse Events by System

  Organ Class and Preferred Term

  Organ Class and

  - (9) Treatment-Emergent Adverse Events by System Organ Class and

  - (11) Drug-Related Treatment-Emergent Adverse Events of Clinical Interest by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

### Number of subjects

- Summary tables other than (5), (6) and (9) A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.
- Summary tables for (5) and (6) A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.
- Summary table for (9) A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT. When calculating percentages for each time interval, the number of subjects at risk (i.e., subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

#### 6.7.2 **Clinical Laboratory Evaluations**

6.7.2.1 Laboratory Tests other than Urinalysis

Analysis Set: Safety Analysis Set Analysis Endpoint(s): See Section 9.3.6.

Using the (Baseline to post Baseline visits) of the visit window

Analytical Method(s): For each endpoint, summaries (1) to (3) will be provided.

(1) Summary of Laborator T (1) Summary of Laboratory Test Results and Change from Baseline

Descriptive statistics for observed values and changes from

Kerms of Use baseline (each post-baseline visit - Baseline) will be provided by subject type for each visit.

(2) Case Plots Plots over time for each subject will be presented.

(3) Summary of Shifts of Laboratory Test Results Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided by subject type.

For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

ld subject

#### 6.7.2.2 Urinalysis

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): See Section 9.3.6.

Using the (Baseline to post Baseline visits) of the visit window Visit:

defined in Section 9.2.2

Analytical Method(s): For pH and specific gravity, summaries (1), (2) and (4) will be

provided.

type.

For each endpoint other than pH and specific gravity, summaries (3) and (4) will be provided.

(1) Summary of Urine Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided by subject type for each visit.

(2) Case Plots Plots over time for each subject will be presented.

Property of Takeda. For non's (3) Number of Subjects in Categories of Urine Laboratory Test Results Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided by subject

(4) Summary of Shifts of Urine Laboratory Test Results Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided by subject type.

Diastolic Blood Pressure

Body Temperature

leight
espir For each urine laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

#### 6.7.3 Vital Signs, Weight and Height

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): Systolic Blood Pressure

Heart Rate

Weight

Respiration Rate **BMI** 

Using the (Baseline to post Baseline visits) of the visit window Visit:

defined in Section 9.2.2.

Analytical Method(s): For each endpoint, summaries (1) and (2) will be provided.

(1) Summary of Vital Signs, Weight and Height, and Change from

Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided by

subject type for each visit.

(2) Case Plots

Plots over time for each subject will be presented.

#### 6.7.4 **ECGs**

Safety Analysis Set Analysis Set:

point, of takeda. Analysis Endpoint(s): Heart Rate

RR Interval PR Interval **QRS** Interval QT Interval **QTcF** Interval

Interpretation [Within Normal Limits, Abnormal but not

Clinically Significant, Abnormal and

Clinically Significant]

Visit: Using the (Baseline to post Baseline visits) of the visit window

defined in Section 9.2.2.

Analytical Method(s): For each endpoint other than 12-lead ECG interpretations, summaries

(1) and (2) will be provided.

For ECG interpretation, summary (3) will be provided.

(1) Summary of ECG Parameters and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided by subject type for each visit.

(2) Case Plots
Plots over time for each subject will be presented.

(3) Summary of Shift of ECG Interpretation
Shift table showing the number of subjects in each category at baseline and each post-baseline visit will be provided by subject type.

# 6.7.5 Displays of Treatment-Emergent Adverse Events (Japanese)

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): TEAE

Analytical Method(s): TEAEs will be summarized in the same way as in Section 6.7.1.2. All

summaries will be presented in Japanese.

### 6.8 Pharmacokinetic, Pharmacodynamic, and Biomarker Analyses

### 6.8.1 Pharmacokinetic Analysis

Not applicable.

### 7.0 REFERENCES

[1] World Health Organization (WHO) growth charts "A SAS Program for the WHO Growth Charts (ages 0 to <2 years)"

https://www.cdc.gov/nccdphp/dnpao/growthcharts/resources/sas-who.htm

[2] Centers for Disease Control (CDC) growth charts "A SAS Program for the 2000 CDC Growth Charts (ages 0 to <20 years)"

https://www.cdc.gov/nccdphp/dnpao/growthcharts/resources/sas.htm

### 8.0 CHANGES TO PROTOCOL PLANNED ANALYSES

There was no change to the protocol planned analyses.

#### 9.0 **APPENDIX**

#### 9.1 **Changes From the Previous Version of the SAP**

Not applicable.

#### 9.2 **Data Handling Conventions**

#### 9.2.1 **Definition of Study Days**

The following definitions and calculation formulas will be used.

- phicable Terms of Use Study Day: The day before the first dose of the study drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. If the date of the observation is on the same date or after the day of the first dose, Study Day will be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.
- Follow-up Day: The day after the last dose of the study drug will be defined as Follow-up Day 1.

#### **Definition of Study Visit Windows** 9.2.2

When calculating Study Day relative to a reference date (ie, date of first dose of study drug [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0.

When calculating Follow-up Day relative to a reference date (ie, date of last dose of study drug [Follow-up Day 0]), it will be calculated as: date of observation - reference date. Hence, reference day is always Follow-up Day 0.

All evaluable data (ie, non-missing data) will be handled according to the following rules.

### Endpoints other than ItchRO Scores and PK Samples 9.2.2.1

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used. For laboratory test data, if there are two observations of both central laboratory sample and local sample on the same date, central laboratory sample data will be used. Values less than or equal to the lower limit of quantification will be treated as one-half of the lower limit value when calculating the descriptive statistics. Values greater than or equal to the upper limit of quantification will be treated as the upper limit value when calculating the descriptive statistics.

Table 9.1 Visit Window of sBA

| | Scheduled Study Day<br>(days) | | Time Interval (days) | |
|---|---|---|---|---|
| Visit | | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: | 1 | -42 - 1 | 10) |
| Week 12 | Study Day: | 85 | 2 - 106 | <15 |
| Week 18 | Study Day: | 127 | 107 - 141 | <b>≥</b> 15 |
| Week 22 | Study Day: | 155 | 142 - 169 | <15 |
| Week 28 | Study Day: | 197 | 170 - 232 | <15 |
| Week 38 | Study Day: | 267 | 233 - 302 | <15 |
| Week 48 | Study Day: | 337 | 303 - 379 | <15 |
| Week 18 (LOCF) | Study Day: | 127 | 2 - 141 | <15 |
| Week (48 + 12 * n) (n=1, 2,) | Study Day: | 337 + 12 * 7 * (n) | (337 + 12 * 7 * (n) -<br>41) - (337 + 12 * 7 *<br>(n) + 42) | < 15 |

Table 9.2 Visit Window of Liver Enzymes (ALT, ALP) and Bilirubins (Total and Direct)

| | Scheduled Study Day<br>(days) | | Time Interval (days) | |
|---|---|---|---|---|
| Visit | | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: | 1 | -42 - 1 | |
| Week 3 | Study Day: | 22 | 2 - 32 | <15 |
| Week 6 | Study Day: | 43 | 33 - 64 | <15 |
| Week 12 | Study Day: | 85 | 65 - 106 | <15 |
| Week 18 | Study Day: | 127 | 107 - 141 | <15 |
| Week 22 | Study Day: | 155 | 142 - 169 | <15 |
| Week 28 | Study Day: | 197 | 170 - 232 | <15 |
| Week 38 | Study Day: | 267 | 233 - 302 | <15 |
| Week 48 | Study Day: | 337 | 303 - 379 | <15 |
| Week 18 (LOCF) | Study Day: | 127 | 2 - 141 | <15 |
| Week (48 + 12 * n) (n=1, 2,) | Study Day: | 337 + 12 *<br>7 * (n) | (337 + 12 * 7 * (n) -<br>41) - (337 + 12 * 7 *<br>(n) + 42) | < 15 |

Visit Window of Vital Signs, Weight and Height, Table 9.3 , CBC, Coagulation, Chemistry Panel,

**Urinalysis, Serum Storage Samples** 

| | Scheduled Study Day<br>(days) | | Time Interval (days) | |
|---|---|---|---|---|
| Visit | | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: | 1 | -42 - 1 | 2/6 |
| Week 3 | Study Day: | 22 | 2 - 32 | <15 |
| Week 6 | Study Day: | 43 | 33 - 64 | <15 |
| Week 12 | Study Day: | 85 | 65 - 106 | <15 |
| Week 18 | Study Day: | 127 | 107 - 141 | <15 |
| Week 22 | Study Day: | 155 | 142 - 176 | <15 |
| Week 28 | Study Day: | 197 | 177 - 232 | <15 |
| Week 38 | Study Day: | 267 | 233 - 302 | <15 |
| Week 48 | Study Day: | 337 | 303 - 379 | <15 |
| Week (48 + 12 * n) (n=1, 2,) | Study Day: | 337 + 12 *<br>7 * (n) | (337 + 12 * 7 * (n) -<br>41) - (337 + 12 * 7 *<br>(n) + 42) | < 15 |

Table 9.4

| Visit | Scheduled St<br>(days | | Time Interv | Follow-up Da |
|---|---|---|---|---|
| Baseline (Week 0) | Study Day: | 1 | -42 - 1 | |
| Week 12 | Study Day: | 85 | 2 - 141 | <15 |
| Week 28 | Study Day: | 197 | 142 - 267 | <15 |
| Week 48 | Study Day: | 337 | 268 - 379 | <15 |
| Week (48 + 12 * n) (n=1,2,) | Study Day: | 337 + 12 * 7 * (n) | (337 + 12 * 7 * (n) -<br>41) - (337 + 12 * 7 *<br>(n) + 42) | < 15 |
| 3 of Takeda. | | | | |



Table 9.7 Visit Window of Lipid Panel, Cholestasis Biomarkers (sBA subspecies, C4, FGF19, Autotaxin), Lipid Soluble Vitamins

| | Scheduled Study Day<br>(days) | | Time Interval (days) | |
|---|---|---|---|---|
| Visit | | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: | 1 | -42 - 1 | |
| Week 12 | Study Day: | 85 | 2 - 106 | <15 |
| Week 18 | Study Day: | 127 | 107 - 141 | <15 |
| Week 22 | Study Day: | 155 | 142 - 169 | <15 |
| Week 28 | Study Day: | 197 | 170 - 232 | <15 |
| Week 38 | Study Day: | 267 | 233 - 302 | <15 |
| Week 48 | Study Day: | 337 | 303 - 379 | <15 |
| Week (48 + 12 * n) (n=1, 2,) | Study Day: | 337 + 12 *<br>7 * (n) | (337 + 12 * 7 * (n) -<br>41) - (337 + 12 * 7 *<br>(n) + 42) | < 15 |

#### 9.2.2.2 PK Samples

Not applicable.

#### 9.2.2.3 ItchRO Weekly Average Scores

ms of Use For visits other than Week 18 (LOCF), weekly average scores are calculated as the average of the scores (morning, evening, daily average of morning and evening, or daily maximum of morning and evening) over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). For the change from baseline calculations in weekly average ItchRO scores, baseline is defined in Table 9.8. Post-baseline weekly average ItchRO scores are only computed if at least 4 of the 7 daily ItchRO scores for the 7-day period are available. The restriction is not set for baseline ItchRO average

In the event that a subject/caregiver failed to complete the morning/evening report, the morning/evening score for that day will be treated as missing data.

For Week 18 (LOCF), if a subject/caregiver is not compliant with reporting ItchRO assessments during the 7-day period on or before the visit, the weekly average score from the most recent, previous compliant 7-day period will be used in a LOCF format. This process will be repeated as necessary. For example, if the 7-day period on or before the Week 18 (LOCF) visit (e.g., Study Days 120-126) is non-compliant, then Study Days 113-119 would be used.

Visit Window of ItchRQ Weekly Average Score Table 9.8

| | Scheduled Study Day<br>(days) | | Time Interval (days) | |
|---|---|---|---|---|
| Visit | | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: | -1 | -71 | |
| Week 3 | Study Day: | 21 | 15 - 21 | <15 |
| Week 6 | Study Day: | 42 | 36 - 42 | <15 |
| Week 12 | Study Day: | 84 | 78 - 84 | <15 |
| Week 18 | Study Day: | 126 | 120 - 126 | <15 |
| Week 19 | Study Day: | 133 | 127 - 133 | <15 |
| Week 20 | Study Day: | 140 | 134 - 140 | <15 |
| Week 21 | Study Day: | 147 | 141 - 147 | <15 |
| Week 22 | Study Day: | 154 | 148 - 154 | <15 |
| Week 28 | Study Day: | 197 | 191 - 197 | <15 |
| Week 38 | Study Day: | 267 | 261 - 267 | <15 |
| Week 48 | Study Day: | 337 | 331 - 337 | <15 |
| Week 18 (for LOCF and | Study Day: | 126 | 1 - 126 | <15 |
| Week (48 + 12 * n) (n=1, 2,) | Study Day: | 337 + 12 * 7 * (n) | (337 + 12 * 7 * (n) -<br>6) - (337 + 12 * 7 *<br>(n)) | < 15 |

#### 9.2.3 **Partial Date Conventions**

For Medication History and Concomitant Medication, if their stop date is partially/completely missing, following handling rules will be applied.

```
3ct to the applicable Terms of Use
if (CMCAT="MEDICATION HISTORY") then "(1) Medical History";
else if (CMENRTPT="ONGOING") then "(3) Concomitant Medication";
else if
(. < medication end year < TAK-625 start year) or
    medication end year = TAK-625 start year and
 . < medication end month < TAK-625 start month) or
    medication end year = TAK-625 start year and
    medication end month = TAK-625 start month and
 else "(3) Concomitant Medication";
```

#### 9.3 **Derivation of Endpoints**

### Change from Week 18 to Week 22 of Primary and Secondary Efficacy Endpoints 9.3.1

For each endpoint (primary and secondary efficacy endpoints), the change from Week 18 to Week 22 of the endpoint is defined as the difference between a value at Week 22 and a value at Week 18 (LOCF).

#### 9.3.2 **ItchRO** Average Scores

Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) or more frequent (Item 3) itching.

ItchRO(Obs/Pt) Weekly Average Morning Score: Sum of ItchRO daily morning scores (over a 7-day period) divided by the number of days ItchRO completed. The definition applies to both severity (Item 1) weekly average scores.

ItchRO(Obs/Pt) Weekly Average Severity Score (based on the daily maximum of morning and evening scores): Sum of ItchRO(Obs) daily maximum of morning and evening scores (over a 7-day period) divided by the number of days ItchRO completed.

- ItchRO (Obs/Pt) Weekly Average Severity Score (based on the daily average of morning and evening scores): Sum of ItchRO(Obs) daily average of morning and evening scores (over a 7-day period) divided by the number of days ItchRO completed.
- ItchRO(Obs/Pt) 4-Week Average Morning Score: Sum of ItchRO daily morning scores (over a 28-day period) divided by the number of days ItchRO completed. The definition applies to both severity (Item 1) and frequency (Item 3, Observer only) 4-week average scores.
- ItchRO(Obs/Pt) 4-Week Average Evening Score: Sum of ItchRO daily evening scores (over a 28-day period) divided by the number of days ItchRO completed. The definition applies to both severity (Item 1) and frequency (Item 3, Observer only) 4-week average scores.




# **9.3.5 Z-scores**

Z-scores of weight, height and BMI are based on a subject's gender and age at each scheduled visit. For subjects less than 24 months of age, the World Health Organization (WHO) growth charts are recommended by the Centers for Disease Control (CDC) and will be used to derive z-scores. For subjects at least 24 months of age, the CDC growth charts will be used to derive z-scores.

Age at which height and weight were measured should be used for calculating z-scores, not using age at baseline.

# 9.3.6 Lists of Laboratory Tests

| | ratory rests | | 0, |
|---|---|---|---|
| Hematology (CBC with | <b>Chemistry</b> | Lipid Panel | <u>Urinalysis</u> |
| <u>Differential)</u> | Albumin | Total cholesterol | pН |
| Hematocrit | ALP | LDL-C (direct) | Specific gravity |
| Hemoglobin | Amylase | HDL-C | Protein |
| MCV, MCH, MCHC | ALT (SGPT) | TG (V) | Glucose |
| Red blood cells | AST (SGOT) | 250 | Ketones |
| Platelets | Bicarbonate | Cholestasis Biomarkersa | Bilirubin |
| White blood cells | Bilirubin, direct | sBA (LC-MS) | Occult blood and cells |
| WBC Differential (% and | (conjugated) | sBA subspecies | Nitrite |
| absolute) | Total serum Bilirubin | 7alpha-hydroxy-4- | Urobilinogen |
| Neutrophils | (TSB) | cholesten-3-one (C4) | Leukocyte esterase |
| Eosinophils | BUN | FGF-19 | Microscopic examination |
| Basophils | Calcium | Autotaxin | Oxalate |
| Lymphocytes | Chloride | | Urinary creatinine |
| Monocytes | Creatinine | Lipid Soluble | , |
| | GGTO | <u>Vitamins</u> | Marker of HCC |
| <b>Coagulation</b> | Glucose | 25-hydroxy vitamin D | AFP |
| aPTT (sec) | Lipase | Retinol | 1111 |
| INR | Phosphate | RBP | |
| PT (sec) | Potassium | Alpha-tocopherol | |
| 70. | Sodium | Estimated Total Lipids | |
| 100 | Corrected Sodium | Ratio of Alpha-tocopherol | |
| 101 | Total protein | to Estimated Total Lipids | |
| aPTT (sec) INR PT (sec) | Total sBA (enzymatic assay) | | |
| 77 | Uric Acid | | |
| | Measured serum<br>Osmolality | | |

# Property of Takeda: For non commercial use only and subject to the applicable Terms of tuse

Properly of Takeda: For non-commercial use only and subject to the applicable Terms



Study Number: TAK-625-3001

Open-Label, Phase 3 Study to Evaluate the Efficacy and Safety of TAK-625 in the Treatment of Subjects with Alagille Syndrome
Phase: 3
Version: 2.0
Date: 10-Nov-2023

Prepared by:

Based on:
Protocol Version: Amendment 2
Protocol Date: 08-Dec-2022

Protocol Date: 08-Dec-2022

Protocol Date: 07-Dec-2022

Protocol Date: 08-Dec-2022

Protocol Date: 08-Dec-2022

Protocol Date: 08-Dec-2022

# **REVISION HISTORY**

| 1.0 01-Jul-2022 Not Applicable 2.0 See Section 9.1 | |
|---|---|
| See Section 9.1 See Section 9.1 | See Section 9.1 See Section 9.1 The application of the application o |
| ise only and siliplect to | non-commercial use only and subject to |
| | , non-commercial c |

# TABLE OF CONTENTS

| 1.0 | | OBJEC | TIVES, ENDPOINTS AND ESTIMANDS | 9 |
|---|---|---|---|---|
| | 1.1 | | ectives | |
| | | 1.1.1 | Primary Objective | |
| | | 1.1.2 | Primary Objective Secondary Objective(s) | ( <u>(</u> ) |
| | | 1.1.3 | Additional Objective(s) | 9 |
| | 1.2 | Enc | lpoints | 9 |
| | | 1.2.1 | Additional Objective(s) Ipoints Primary Endpoint(s) Secondary Endpoint(s) 2.1 Key Secondary Endpoints(s) | 9 |
| | | 1.2.2 | Secondary Endpoint(s) | 9 |
| | | 1.2. | 2.1 Key Secondary Endpoints(s) | 9 |
| | | 1.2. | 2.2 Secondary Endpoint(s) | 9 |
| | | 1.2.4 | Safety Endpoints | 11 |
| | | 1.2.5 | Other Endpoints | 11 |
| | | 1.2. | Safety Endpoints Other Endpoints 5.1 PK Endpoint imand(s) Y DESIGN | 11 |
| | 1.3 | Esti | imand(s) | 11 |
| 2.0 | | STUDY | Y DESIGN | 11 |
| 3.0 | | STATIS | STICAL HYPOTHESES AND DECISION RULES | 13 |
| 4.0 | | SAMPI | LE-SIZE DETERMINATION | 13 |
| 5.0 | | | YSIS SETS | |
| | 5.1 | | Subjects Who Signed the Informed Consent Form | |
| | 5.2 | | Subjects Who Did Not Enter the Treatment Period | |
| | 5.3 | | ety Analysis Set | |
| | 5.4 | | ention-to-treat set (ITT) | |
| | 5.5 | | dified Intention-to-treat set (MITT) | |
| <i>(</i> 0 | 5.6 | | -Protocol Analysis Set (PPS) | |
| 6.0 | | ~ 0. | STICAL ANALYSIS | |
| | 6.1 | Ger | neral Considerations | |
| | 6.2 | | alysis Approach | |
| 4 | 0 | 6.2.1 | Analysis Approach for Continuous Efficacy Endpoints | |
| | | 6.2.2<br>6.2.3 | Analysis Approach for Binary Efficacy Endpoints | |
| | 6.3 | | Analysis Approach for Time-to-Event Efficacy Endpoints position of Subjects | |
| | 0.3 | 6.3.1 | Study Information | |
| | | 632 | Screen Failures | 10<br>18 |

| | 6.3.3 | Sub | ject Eligibility | 18 |
|---|---|---|---|---|
| | 6.3.4 | | nber of Subjects Who Entered the Treatment Period by Site | |
| | 6.3.5 | Disp | cocol Deviations and Analysis Sets | 19 |
| | 6.3.6 | Prot | tocol Deviations and Analysis Sets | 20 |
| | 6.3. | 6.1 | Significant Protocol Deviations | 20 |
| | 6.3. | 6.2 | Analysis Sets | 20 |
| 6.4 | Der | nogra | phic and Other Baseline Characteristics | 21 |
| | 6.4.1 | Den | nographic and Baseline Characteristics | 21 |
| | 6.4.2 | Med | Analysis Sets | 24 |
| 6.5 | Med | dicatio | on History and Concomitant Medications | 24 |
| 6.6 | Ext | ent of | Exposure and Compliance | 25 |
| 6.7 | Effi | cacy | Analysis | 25 |
| | 6.7.1 | Prin | Analysis | 25 |
| | 6.7. | 1.1 | Primary Analysis | 25 |
| | 6.7. | 1.2 | Sensitivity Analysis | 25 |
| | 6.7.2 | Seco | ondary Endpoints Analysis | 26 |
| | 6.7. | 2.1 | Key Secondary Endpoints | 26 |
| | 6.7. | 2.2 | Sensitivity Analysis | 20 |
| | 6.7. | 2.3 | Secondary Endpoints | 27 |
| | 6.7.4 | Sub | group Analysis | 30 |
| 6.8 | Safe | ety Aı | group Analysisalysisverse Events | 31 |
| | 6.8.1 | Adv | verse Events | 31 |
| | 6.8. | 1.1 | Overview of Treatment-Emergent Adverse Events | 31 |
| , 1 | 6.8. | 1.2 | Displays of Treatment-Emergent Adverse events | 32 |
| OX | 6.8. | 1.3 | Displays of Pretreatment Events | 34 |
| } | 6.8.2 | Clin | ical Laboratory Evaluations | 34 |
| | 6.8. | 2.1 | Laboratory Tests other than Urinalysis | 34 |
| | 6.8. | 2.2 | Urinalysis | 35 |
| | 6.8.3 | Vita | ıl Signs, Weight and Height | 36 |
| | 6.8.4 | ECC | Gs | 36 |

| | 6.8.5 | Displays of Treatment-Emergent Adverse Events (Japanese) | 37 |
|---|---|---|---|
| 6.9 | Ph | armacokinetic, Pharmacodynamic, and Biomarker Analyses | 37 |
| | 6.9.1 | Pharmacokinetic Analysis | 37 |
| | | Pharmacokinetic Analysis | 37 |
| 7.0 | REFEI | RENCES | 38 |
| 8.0 | CHAN | GES TO PROTOCOL PLANNED ANALYSES | 38 |
| 9.0 | APPE | NDIX | 38 |
| 9.1 | Ch | NDIX | 38 |
| 9.2 | Da | ta Handling Conventions | 50 |
| | 9.2.1 | Definition of Study Days | 50 |
| | 9.2.2 | Definition of Study Visit Windows | 50 |
| | 9.2 | .2.1 Endpoints other than ItchRO Scores and PK Samples | 50 |
| | 9.2 | .2.2 PK Samples | 53 |
| | 9.2 | .2.3 ItchRO Weekly Average Scores | 53 |
| | 9.2 | 2.4 ItchRO 4-week Average Scores Partial Date Conventions rivation of Endpoints Change from Week 18 to Week 22 of Primery and Secondary Efficiency | 54 |
| | 9.2.3 | Partial Date Conventions | 55 |
| 9.3 | De | rivation of Endpoints | 55 |
| | 9.3.1 | Change from Week 18 to Week 22 of Primary and Secondary Efficacy Endpoints | |
| | | Endpoints | 55 |
| | 9.3.2 | ItchRO Average Scores | 56 |
| | 9.3.5 | Z-scores | |
| | 9.3.6 | Lists of Laboratory Tests | |
| | 9.3.7 | Table for AECI | |
| | 9.3.8 | Significance Level and Confidence Coefficient | |
| 9.4 | - An | alysis Software | 59 |
| | An | | |
| LIST | OF IN- | TEXT TABLES | |
| Table 9 | 9.1 | Visit Window of sBA | 51 |
| Table 9 | 9.2 | Visit Window of Liver Enzymes (ALT, ALP) and Bilirubins (Total and | |
| | | Direct) | 51 |
| Table 9 | 9.3 | Visit Window of Vital Signs, Weight and Height, | |
| | | Urinalysis, Serum Storage Samples | <b>5</b> 1 |
| | | Official solution of the contract of the contr | ·····J |

| 1 autc 9.5 | Visit Window of ECGs |
|---|---|
| Table 9.8 | Visit Window of Lipid Panel, Cholestasis Biomarkers (sBA subspecies FGF19), Lipid Soluble Vitamins |
| Table 9.9 | Visit Window of PK |
| Table 9.10 | Visit Window of ItchRO Weekly Average Score |
| Table 9.11 | Visit Window of ItchRO 4-week Average Score |
| | ×O |
| LIST OF IN | N-TEXT FIGURES |
| Figure 2.1 | Schematic Study Design |
| | 35 |
| | allo |
| | th. |
| | N <sub>S</sub> S |
| | ial use |
| | ercialuse |
| | mnercialuse |
| | commercial use |
| | on commercial use |
| | or non-commercial use |
| | . For non-commercial use |
| | da. For non-commercial use |
| | da: For non-commercial use |
| x x x e | da. For non-commercial use |
| etate | da. For non-commercial lise |
| it of de | da. For non-commercial use |
| it of take | Visit Window of Lipid Panel, Cholestasis Biomarkers (sBA subspecies FGF19), Lipid Soluble Vitamins Visit Window of PK |

### **ABBREVIATIONS**

ΑE adverse event

**AECI** adverse event of clinical interest

AFP alpha-fetoprotein **ALGS** Alagille syndrome ALP alkaline phosphatase **ALT** alanine aminotransferase analysis of covariance ANCOVA

aPTT activated partial thromboplastin time

AST aspartate aminotransferase 7αC4 7α-hydroxy-4-cholesten-3-one

BMI body mass index **BUN** blood urea nitrogen **CBC** complete blood count CI confidence interval

Electrocardiogram **ECG** 

fibroblast growth factor 19 FGF-19

gamma-glutamy/transferase **GGT** hepatocellular carcinoma **HCC** 

high density lipoprotein-cholesterol HDL-C

health-related quality of life HRQoL

ItchRO Observer ItchRO(Obs) ItchRO(Pt) ItchRO Patient

ITT intention-to-treat set

KM Kaplan-Meier

LDT-C low density lipoprotein-cholesterol

LIN lower limit of normal

last observation carried forward

Proper Is LS means least square means lipid soluble vitamin

MCH mean corpuscular hemoglobin

**MCHC** mean corpuscular hemoglobin concentration

Medical Dictionary for Regulatory Activities MedDRA

MITT modified intention-to-treat set **PEBD** partial external biliary diversion

pharmacokinetic PK

**PPS** per-protocol analysis set PRO patient-reported outcomes

PT preferred term 25th percentile Q1 75th percentile Q3

QT interval corrected using Bazett's formula QTcB QTcF QT interval corrected using Fridericia's formula only and suf

quality-of-life QOL

RBP retinol binding protein serious adverse event SAE SAP statistical analysis plan

serum bile acid sBA

serum bile acid serum glutamic-oxaloacetic transaminase **SGOT** serum glutamic-pyruvic transaminase **SGPT** 

SOC system organ class

TEAE treatment-emergent adverse event

triglycerides TG

WBC
WHODrug total serum bilirubin upper limit of normal white blood cell

World Health Organization Drug Dictionary

### 1.0

# 1.1

# 1.1.1

# 1.1.2

- To evaluate the PK of TAK-625 in subjects with ALGS.

  To evaluate the efficacy of TAK-625 on biochemical markers of cholestasis and liver disease in subjects with ALGS.

  Additional Objective(s)

  Applicable

  Endpoints

  Primary Endpoint\*\*

# 1.1.3

Not Applicable

### 1.2

# 1.2.1

The change from Week 18 to 22 of fasting sBA levels.

### Secondary Endpoint(s) 1.2.2

### Key Secondary Endpoints(s) 1.2.2.1

- Change from baseline to Week 18:
  - *♦ Fasting sBA levels.*
  - ♦ Pruritus as measured by ItchRO (Obs): weekly average severity (based on daily maximum of morning and evening severity scores).
  - ♦ Pruritus as measured by ItchRO (Obs): weekly average morning severity.
- Change from Week 18 to 22:
  - Pruritus as measured by ItchRO (Obs): weekly average severity (based on daily maximum of morning and evening severity scores).
  - Pruritus as measured by ItchRO (Obs): weekly average morning severity.

### Secondary Endpoint(s)

- Change from baseline to Week 18:
  - Pruritus as measured by Patient-reported Itch Reported Outcome (ItchRO [Pt]): weekly average severity (based on daily maximum of morning and evening severity scores).



### 1.2.4 **Safety Endpoints**

Incidence of AEs including SAEs, related to study drug, leading to study drug discontinuation, and AEs of clinical interest (AECIs).

AECIs include the following:

- *♦ LSV deficiency events.*
- Liver parameter disruption.
- 3ble Terms of Use Change from baseline in clinical laboratory values (hematology, chemistry, urinalysis, and others), physical examination findings (including body weight, height, and body mass index [BMI]), vital signs, and electrocardiogram (ECG) parameters.

### 1.2.5 **Other Endpoints**

### 1.2.5.1 PK Endpoint

- Plasma levels of TAK-625 at predose and approximately 4 hours after the morning dose at Week 12.
- Plasma levels of TAK-625 at predose (optional) and approximately 30 minutes after morning Plasma levels of 1AA-025 at product dose at Week 18 (or any visit up to Week 28).

### Estimand(s) 1.3

Not Applicable.

### 2.0 STUDY DESIGN

This is a phase 3, multicenter, open-label, uncontrolled study to evaluate the efficacy and safety of TAK-625 in the treatment of Japanese subjects with ALGS.

# Study Population:

The study population is defined as "Japanese patients with ALGS who are 1 year of age or older".

Study Period Screening, Treatment [Dose Escalation, Stable Dosing, and Follow-up Dosing], and Safety Follow-up Period):

This study consists of the screening period (up to 6 weeks prior to the study administration), 2-week dose escalation period (doses up to 400 µg/kg/day, once a day [OD], as tolerated), 46-week stable dosing period, and follow-up dosing period (until TAK-625 is approved or available in Japan commercially, or if the subject withdraws from the study, or if the investigator determines the subject's discontinuation, or if the sponsor stops the program or development in this indication).

# 1. Screening Period (Up to 6 Weeks prior to the Study Administration):

In the screening period, for subjects who do not have documentation of mutation related to ALGS (JAGGED-1 or NOTCH2), genetic testing may be performed, if necessary. The electronic diary (eDiary) for assessing pruritus with the Itch Reported Outcome (ItchRO) instrument will be dispensed and subjects and caregivers will undergo training during the screening visit.

# 2. <u>Dose Escalation Period (2 Weeks: Week 0 to 2):</u>

In the 2-week dose escalation period, at the baseline visit (Week 0/Visit 2), subjects will be assessed to confirm continued study eligibility and undergo a physical examination including body weight, height, BMI, and vital signs, and have urine and blood samples taken for hematology, chemistry, fasting lipid panel, baseline levels of sBA, and other cholestasis biochemical markers. Compliance with ItchRO will be assessed. Study drug for Weeks 1 and 2 will be supplied at the baseline visit to eligible subjects. Subjects will receive the study drug, TAK-625, administered orally OD. The dose will be increased weekly over a 2-week period up to 400 μg/kg/day QD as follows: dose level 1, 200 μg/kg/day QD for 1 week; and dose level 2, 400 ug/kg/day OD for the remaining duration of the study. If an individual subject exhibits a treatment-emergent moderate or severe drug-related gastrointestinal (GI) toxicity with 400 μg/kg/day, study drug dose may be lowered to 200 μg/kg/day; later attempts to escalate the dose are permitted during the dose escalation period. This decision should be made in consultation with the medical monitor. If further dose escalations fail during the dose escalation period, the subject will remain on 200 μg/kg/day for the remainder of the study. The dose should be taken at least 30 minutes prior to the first meal of the day. It is recommended that the dose should be taken approximately at the same time each day for the duration of the treatment period. Subjects will return to the clinic at Week 3 and follow-up phone calls will be made at Weeks 1 and 2.

# 3. Stable Dosing Period (46 Weeks: Week 3 to 48):

After the dose escalation period, each subject will continue dosing with study drug at the Week 3 dose level, which is either 200 or 400 µg/kg/day, in the stable dosing period. Subjects will visit the study site at Weeks 6, 12, 18, 22, 28, 38, and 48, and undergo physical examinations. Subject contacts (phone calls) will be conducted as appropriate throughout the stable dosing period. Subjects and caregivers will continue twice daily completion of their ItchRO throughout the period.

# 4. Follow-up Dosing Period (after Week 48):

In the follow-up dosing period, each subject will continue dosing with study drug at the Week 48 dose level, which is either 200 or 400 µg/kg/day. The safety evaluation will be performed in all the subjects every 12 weeks from Week 48 visit until TAK-625 is approved or available in Japan commercially, or if the subject withdraws from the study, or if the investigator determines the subject's discontinuation, or if the sponsor stops the program or development in this indication. Bile acids and ItchRO will be measured to evaluate the long-term effectiveness of TAK-625. For subjects discontinuing early, safety follow-up will be conducted.

# 5. Safety Follow-up (after Final Visit/Early Termination [ET]):

Subjects/caregivers will have a final safety follow-up subject contact (phone call) 7 days after the final study visit or ET visit (except for screen failure).

A schematic of the study design is included as Figure 2.1.

**Schematic Study Design** Figure 2.1



### STATISTICAL HYPOTHESES AND DECISION RULES 3.0

Not Applicable.

### SAMPLE-SIZE DETERMINATION 4.0

ALGS is a rare disease. The targeted sample size is approximately 5 subjects based on enrollment feasibility of this population in Japan, rather than power calculation.

### 5.0 **ANALYSIS SETS**

### All Subjects Who Signed the Informed Consent Form 5.1

All subjects who signed the informed consent form.

# All Subjects Who Did Not Enter the Treatment Period

All subjects who did not enter the treatment period.

# Safety Analysis Set

All subjects who received at least one dose of study drug.

# 5.4 Intention-to-treat set (ITT)

All subjects who received at least one dose of study drug.

# 5.5 Modified Intention-to-treat set (MITT)

All subjects who received study drug through Week 18, and had a reduction from baseline in sBA levels of  $\geq$ 50% at the Week 12 or Week 18 measurement.

# 5.6 Per-Protocol Analysis Set (PPS)

All ITT subjects who did not have any of the following major protocol deviations and whose primary endpoint was evaluable.

- Subjects who did not meet inclusion criteria #3, 4, 6, or 10.
- Subjects who met exclusion *criteria* #2, 3, 4, 5, 6, 7, 14, 15, or 16.

### 6.0 STATISTICAL ANALYSIS

Statistical analyses will be performed using all subjects' data up to Week 22 (i.e., up to Day 169 or 25OCT2023) after the data are locked. PK analysis will be performed using all subjects' data up to Week 12 after the data are locked.

### 6.1 General Considerations

The following definitions and calculation formulas will be used.

- Treatment-emergent adverse event (TEAE): An adverse event whose date of onset occurs on or *after* the start of study drug. TEAEs whose date of onset occurred on or before Week 22 visit (ie, the latest visit by Day 169), will be summarized.
- **Pretreatment event (PTE)**: Any untoward medical occurrence in a clinical investigation *subject* who has signed informed consent to participate in a study but prior to administration of study drug.
- **Concomitant medication**: Concomitant medications whose start date occurred on or before Week 22 visit (ie, the latest visit by Day 169), will be summarized.
- **Descriptive statistics for endpoints other than PK**: Number of subjects, mean, standard deviation, standard error, maximum, minimum, and quartiles (Q1, median, and Q3).
- **Descriptive statistics for PK**: Number of subjects, mean, standard deviation, maximum, median, and minimum.
- **Duration of exposure to study drug (days)**: {Date of last dose of study drug or Week 22 visit (ie, the latest visit by Day 169) which comes faster date of first dose of study drug} + 1.
- **Duration of study after baseline (days)**: {Date of last visit/contact or Week 22 visit (ie, the latest visit by Day 169) which comes faster date of first dose of study drug} + 1.

- Study drug compliance (%): Number of study drugs taken / duration of exposure to study drug \* 100 (rounded to 1 decimal place).
- **Dose Level (μg/kg)**: Strength of study drug taken (mg) / (last available body weight (kg) prior to or on the day of study drug taken) \* 1000.
- **Dose Level Categories for PK (μg/kg)**: Categorize by following below calculation rule. If Min <= dose level < 300 μg/kg, then dose level category = 200 μg/kg; if 300 μg/kg <= dose level <= Max, then dose level category = 400 μg/kg.
- Total Drug Exposure (μg/kg): Sum of {number of study drugs taken \* dose level received (μg/kg)}.
- **Average Daily Dose (μg/kg/day)**: Total Drug Exposure (μg/kg) / Duration of exposure to study drug (days).
- ItchRO (Obs/Pt) Daily Maximum of Morning and Evening Scores: Maximum of morning and evening severity scores for each day. The morning and evening severity scores of the same day should be used for the calculation. Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) itching.
- ItchRO (Obs/Pt) Daily Average of Morning and Evening Scores: Average of morning and evening severity scores for each day. The morning and evening severity scores of the same day should be used for the calculation. Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) itching.
- **Time to liver-associated events**: PEBD surgery, listing for liver transplantation, liver decompensation [hepatic encephalopathy, variceal bleeding, ascites, and spontaneous bacterial peritonitis] events, hepatocellular carcinoma (HCC), death, and other.
- Estimated Total Lipids (mg/dL): Cholesterol (mg/dL) + Triglycerides (mg/dL).
- Ratio of Alpha-tocopherol to Estimated Total Lipids (mg/g): 1000 \* Alpha-tocopherol (mg/dL) / Estimated Total Lipids (mg/dL). For Alpha-tocopherol concentrations reported as below the minimum quantitation limit, half of the minimum quantitation limit is used in the calculation.
- Corrected Sodium (mEq/L): sodium (mEq/L) + (0.002 \* Triglycerides (mg/dL)).

• Subject Type: [all subjects including ones under 1 year old (overall), 1 year or older].

- Time Since Original Diagnosis of ALGS (months): (date of first dose date of original diagnosis of ALGS + 1) / 30.44.
- **Significant Protocol Deviation**: Deviation defined in the PDMP as "Important PD" whose Severity Classifications is "major" or "critical".

When reporting derived values or parameters, following presenting rules will be applied.

- For sBA, ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.
  - For measures of median and mean, use 3 decimal places.
  - For measures of standard deviation, standard error of the mean and CI, use 4 decimal places.
  - For measures of minimum and maximum values as well as observed value (for Listing), use 2 decimal places.
  - >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
  - For p-values use 3 decimal places.
  - Presentation of p-values display p-values that would round to 0.000 as <0.001.
- Other than sBA, and ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.
  - For measures of median and mean, use 1 decimal place beyond those used for the measurement.
  - For measures of standard deviation, standard error of the mean and CI, use 2 decimal places beyond those used for the measurement.
  - For measures of minimum and maximum values, use the same number of decimal places as those used for the measurement.
  - >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
  - For p-values use 3 decimal places.
  - Presentation of p-values display p-values that would round to 0.000 as <0.001.
  - BMI should be rounded to 1 decimal place for reporting.
  - ➤ Derived questionnaire scores, and other similar efficacy parameters recorded as integers, should be rounded to 1 decimal place for reporting.
  - Averaged lab results (e.g. Diastolic/Systolic Blood Pressure and Pulse [when taken in triplicate]) should be rounded to 1 decimal place for reporting.

# 6.2 Analysis Approach

# 6.2.1 Analysis Approach for Continuous Efficacy Endpoints

For efficacy endpoints, all continuous endpoints in this trial will use the analysis method below unless stated otherwise in the section specific to an endpoint.

- Change from Week 18 to Week 22:
  - → Descriptive statistics and two-sided 95% confidence interval of mean will be provided for observed values (Week 18 (LOCF) and Week 22) and changes from Week 18 (Week 22 Week 18 (LOCF)) by subject type. For endpoint with multiple visits, these will be provided by visit.
- Change from baseline to post-baseline:
  - Descriptive statistics and two-sided 95% confidence interval of mean will be provided for observed *values* (baseline and post-baseline visits) and changes from baseline (each post-baseline visit baseline) by subject type. For endpoint with multiple visits, these will be provided by visit.

# 6.2.2 Analysis Approach for Binary Efficacy Endpoints

For efficacy endpoints, all binary endpoints in this trial will use the analysis method below unless stated otherwise in the section specific to an endpoint.

• Frequency distribution will be provided by visit, with proportion and the two-sided 95% confidence interval by subject type. For endpoint with multiple visits, these will be provided by visit.

# 6.2.3 Analysis Approach for Time-to-Event Efficacy Endpoints

For efficacy endpoints, all time-to-event endpoints in this study will use the analysis method below unless stated otherwise in the section specific to an endpoint.

• The event-free survival rate and the two-sided 95% confidence intervals will be provided using the Kaplan-Meier method. The event-free survival rate will also be plotted. Time to event will be defined as the date of first dose of study drug to the event which comes fastest. For subjects without an event, time to event will be defined as the date of first dose of study drug to the censoring date, which is the date of the last study visit/contact.

### 6.3 **Disposition of Subjects**

### 6.3.1 **Study Information**

All Subjects Who Signed the Informed Consent Form Analysis Set:

Analysis Endpoint(s): Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Dictionary Version WHO Drug Dictionary Version

SAS Version Used for Creating the Datasets

Analytical Method(s): (1) Study Information

Study information shown in the analysis endpoints section will be

provided.

6.3.2 Screen Failures

All Subjects Who Did Not Enter the Treatment Period Analysis Set:

Analysis Endpoint(s): Age (years)

> Gender [Male, Female]

(1) Screen Failures Analytical Method(s):

Frequency distributions for categorical endpoints and descriptive

statistics for continuous endpoints will be provided.

6.3.3 Subject Eligibility

All Subjects Who Signed the Informed Consent Form Analysis Set:

broberty of Lykega. Analysis Endpoint(s): **Eligibility Status** [Eligible for Entrance into the

Treatment Period, Not Eligible for Entrance into the Treatment Period

Primary Reason for Subject

Not Being Eligible

[AE, Screen Failure (Did not meet inclusion criteria or did meet

exclusion criteria), Protocol Deviation, Lost to Follow-up, Pregnancy, Withdrawal by Subject,

Study Terminated by Sponsor, Other]

Analytical Method(s): (1) Eligibility for Entrance into the Treatment Period

icable Terms of Use Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being eligible, the total number of ineligible subjects will be used as the denominator.

### 6.3.4 Number of Subjects Who Entered the Treatment Period by Site

ITT Analysis Set:

Analysis Endpoint(s): Status of Entrance into the [Entered]

**Treatment Period** 

[Site numbers will be used as Site Stratum:

categories]

(1) Number of Subjects Enrolled by Site Analytical Method(s):

Frequency distribution will be provided for each stratum.

### 6.3.5 **Disposition of Subjects**

ITT Analysis Set:

[Ongoing, Completed Study Drug, Analysis Endpoint(s): Study Drug Completion

Status

Prematurely Discontinued Study

Drug]

Reason for Discontinuation

of Study Drug

[AE, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Lack of Efficacy, Other]

Completion Status of All [Ongoing, Completed Study, Planned Study Visits Prematurely Discontinued Study]

Reason for Discontinuation

of Study

[AE, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject,

Study Terminated by Sponsor, Pregnancy, Lack of Efficacy, Other]

Analytical Method(s): (1) Disposition of Subjects

Frequency distributions will be provided by subject type. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the

denominator.

KW2 of Use

### 6.3.6 **Protocol Deviations and Analysis Sets**

6.3.6.1 Significant Protocol Deviations

ITT Analysis Set:

Analysis Endpoint(s): Significant Protocol Deviation [Informed Consent and Process, ©

> Inclusion Criteria, Exclusion Criteria, Concomitant Medication, Laboratory Assessment, Study Procedures (not safety and efficacy related), Safety, Visit Schedule, IP conditions, IP preparation, IP administration, Subject IP Compliance, Efficacy,

Subject Discontinuation,

Administrative, Patient Reported Outcomes, PK/PD, Other Criteria]

Analytical Method(s): (1) Protocol Deviations

Frequency distribution will be provided for each deviation category by subject type. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be

counted only once.

6.3.6.2 Analysis Sets

[Categories are based on the definitions in

Section 5.0]

[Included]

[Included]

[Included]

[Included]

Analysis Sets
ITT

M''

Analysis Analysis Sets

Analysis Sets

Analysis Sets (1) Subjects Excluded from Analysis Sets

Frequency distributions will be provided by subject type. For (1), a subject who has several reasons for exclusion will be counted once in

able Terms of Use each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

### 6.4 **Demographic and Other Baseline Characteristics**

### 6.4.1 **Demographic and Baseline Characteristics**

ITT Analysis Set:

Analysis Endpoint(s): Age (years)

ale only and sulbl [Male, Female] Gender

Height (cm)

Weight (kg)

BMI (kg/m2)

Height z-score

Weight z-score

BMI z-score

[Yes, No, Unknown]

[Yes, No, Unknown]

Additional

Criv [JAGGED1, NOTCH2]

Vascular abnormalities

```
Skeletal abnormalities
```

Ocular abnormalities

Characteristic facial

**Features** 

Used Anything to Treat Itch

in the Past

Type of Therapy Used to

Treat Itch in the Past (multiple count)

Topical

Oral

Other

Specific Therapy Used to

Treat Itch in the Past

Topical Corticosteroids

Topical Calcineurin

**Inhibitors** 

Topical Antihistamines,

Menthol

Capsaicin

Salicylic acid

**Local Anesthetics** 

Androgens

Anticholestatic Agents

Anticonvulsants

Antidepressants

Antihistamines

Anti-Oxidants

**Binding Resins** 

Colchicine

Cannabinoid Agonist

Property of Takeda. For non's

achRO(Obs) Weekly
Morning
Average Severity (Item 1)
Score
chRO(Obs) Weekly
orning
erage Free
e

Score

sBA (LC MS)

Analytical Method(s): (1) Demographics and Baseline Characteristics

Frequency distributions for categorical endpoints and descriptive statistics for continuous endpoints will be provided by subject type.

### 6.4.2 **Medical History and Concurrent Medical Conditions**

ITT Analysis Set:

Analysis Endpoint(s): Medical History

**Concurrent Medical Conditions** 

ierns of Use (1) Medical History by System Organ Class and Preferred Term Analytical Method(s):

> (2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided by subject type. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

### Medication History and Concomitant Medications 6.5

(1) Medication History by Anatomical Therapeutic Chemical Level 2

Ongoing at Baseline as well as Those That Started After Baseline

Medication History by Anatomical Therapeutic Chemical Loand Preferred Medication Name

(2) Concomitant Medications That Started and Stopped Prior to Baseline by Anatomical Therapeutic Chemical Level 2 and Preferred Medication Name

(3) Concomitant Medications That Started Prior to Congoing at Baseline as well as Those The by Anatomical Therapeutic Chemical Chem Frequency distributions will be provided by subject type. WHO Drug dictionary will be used for coding. Summaries will be provided using names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication names will be counted only once

for that preferred medication names. For anatomical therapeutic chemical level 2, same manners in counting frequency.

### 6.6 **Extent of Exposure and Compliance**

Analysis Set: ITT

Analysis Endpoint(s): Duration of Exposure to

Study Drug (days)

Study Drug Compliance (%)

Total Drug Exposure (µg/kg)

Average Daily Dose

(µg/kg/day)

(1) Study Drug Exposure, Compliance, Total Drug Exposure and Analytical Method(s):

Average Daily Dose

Frequency distributions for categorical endpoints and descriptive statistics for continuous endpoints will be provided by subject type.

### 6.7 **Efficacy Analysis**

### Primary Endpoint Analysis 6.7.1

6.7.1.1 Primary Analysis

Analysis Set:

Change from Week 18 to 22 of fasting sBA levels Analysis Endpoint(s):

Analytical Method(s): See Section 6.2.1.

Sensitivity Analysis 6.7.1.2

Analysis Set **MITT** 

**PPS** 

Analytical Method(s): Change from Week 18 to 22 of fasting sBA levels

See Section 6.2.1. For supportive analysis, the same analysis as the

primary analysis will be performed using the MITT and the PPS to

confirm robustness of the results.

# 6.7.2 Secondary Endpoints Analysis

# 6.7.2.1 Key Secondary Endpoints

Analysis Set:

ITT

Analysis Endpoint(s):

- Change from baseline to Week 18:
  - · Fasting sBA levels.
  - Pruritus as measured by ItchRO (Obs): weekly average severity (based on daily maximum of morning and evening severity scores)
  - · Pruritus as measured by ItchRO (Obs): weekly average morning severity
- Change from Week 18 to Week 22:
  - · Pruritus as measured by ItchRO (Obs): weekly average severity (based on daily maximum of morning and evening severity scores)
  - · Pruritus as measured by ItchRO (Obs): weekly average morning severity

Analytical Method(s): See Section 6.2.1.

6.7.2.2 Sensitivity Analysis

Analysis Set:

**PPS** 

Analysis Endpoint(s):

- Change from baseline to Week 18:
  - · Fasting sBA levels.
  - · Pruritus as measured by ItchRO (Obs): weekly average severity (based on daily maximum of morning and evening severity scores)
  - · Pruritus as measured by ItchRO (Obs): weekly average morning severity
- Change from Week 18 to Week 22:
  - Pruritus as measured by ItchRO (Obs): weekly average severity (based on daily maximum of morning and evening severity scores)
  - · Pruritus as measured by ItchRO (Obs): weekly average morning severity

Analytical Method(s):

able rems of Use See Section 6.2.1. For supportive analysis, the same analysis as the previous analysis for the key secondary endpoints will be performed using the PPS to confirm robustness of the results.

### 6.7.2.3 Secondary Endpoints

Analysis Set:

ITT

Analysis Endpoint(s):

- Change from baseline to Week 18:
  - Pruritus as measured by ItchRO (Pt): weekly average severity (based on daily maximum of morning and evening severity scores)
  - · Pruritus as measured by ItchRO (Pt); weekly average morning
  - · Liver enzymes (ALT, ALP) and bilirubin (total and direct)
- Change from Week 18 to Week 22:
  - · Pruritus as measured by ItchRO (Pt): weekly average severity (based on daily maximum of morning and evening severity scores)
  - Pruritus as measured by ItchRO (Pt): weekly average morning severity
  - Liver enzymes (ALT, ALP) and bilirubin (total and direct)

Visit:

Using the (Baseline to Week 22) of the visit window defined in Section 9.2.2.

See Section 6.2.1. Analytical Method(s):





Property of Takeor





# 6.7.4 Subgroup Analysis

Analysis Set:

ITT

Analysis Endpoint(s):

- Change from baseline to Week 18:
  - · Fasting sBA levels.
  - Pruritus as measured by ItchRO (Obs): weekly average severity (based on daily maximum of morning and evening severity scores)
  - Pruritus as measured by ItchRO (Obs): weekly average morning severity
- Change from Week 18 to Week 22:
  - · Fasting sBA levels
  - Pruritus as measured by ItchRO (Obs): weekly average severity (based on daily maximum of morning and evening severity scores)

Pruritus as measured by ItchRO (Obs): weekly average morning severity

Subgroup(s):

Age

 $[Min \le - <7, 7 \le - \le Max]$ 

Gender

[Male, Female]

Analytical Method(s):

Descriptive statistics will be provided for above each subgroup by subject type. The MITT will not be used for the analyses due to small sample size.

### 6.8 **Safety Analysis**

### **Adverse Events** 6.8.1

6.8.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): TEAE

Relationship to Study Drug [Related, Not Related] Categories:

> [Mild, Moderate, Severe] Intensity

The following summaries will be provided by subject type. Analytical Method(s):

(1) Overview of Treatment-Emergent Adverse Events

- 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 2) Relationship of Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
- 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
- Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- Relationship of serious Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
- Property of Takedai. For non-col Serious Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
  - Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below.

# Number of subjects

- Summaries for 2) and 6)
   A subject with occurrences of TEAE in both categories (i.e., Related and Not Related) will be counted once in the Related category.
- Summary for 3)
   A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.
- Summaries other than 2), 3), and 6)
   A subject with multiple occurrences of TEAE will be counted only once.

# Number of events

For each summary, the total number of events will be calculated.

# 6.8.1.2 Displays of Treatment-Emergent Adverse events

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): TEAE

Property of Lakeda. For

Categories: [Mild, Moderate, Severe]

Time of Onset (day) [1-14, 15-Max]

Analytical Method(s): The following summaries will be provided using frequency distribution by subject type.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (8) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (9) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- (10) Treatment-Emergent Adverse Events of Clinical Interest by System Organ Class and Preferred Term
- (11) Drug-Related Treatment-Emergent Adverse Events of Clinical Interest by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

# Number of subjects

- Summary tables other than (5), (6) and (9) A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.
- Summary tables for (5) and (6) A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.
- Property of Takedai. For none Summary table for (9) A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT. When calculating percentages for each time interval, the number of subjects at risk (i.e., subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of
Able Lehms of Use subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

#### 6.8.1.3 Displays of Pretreatment Events

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis Endpoint(s): PTE

The following summaries will be provided using frequency Analytical Method(s):

distribution by subject type.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

(1) Pretreatment Events by System Organ Class and Preferred Term

(2) Serious Pretreatment Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

#### 6.8.2 Clinical Laboratory Evaluations

6.8.2.1 Laboratory Tests other than Urinalysis

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): See Section 9.3.6.

Visit: Using the (Baseline to Week 22) of the visit window defined in

Section 9.2.2.

Analytical Method(s): For each endpoint, summaries (1) to (3) will be provided.

(1) Summary of Laboratory Test Results and Change from Baseline

by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided by

subject type for each visit.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Summary of Shifts of Laboratory Test Results Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided by subject type.

For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be to the applicat based on these classifications.

#### 6.8.2.2 Urinalysis

Analysis Set: Safety Analysis Set

See Section 9.3.6. Analysis Endpoint(s):

Using the (Baseline to Week 22) of the visit window defined in Visit:

Section 9.2.2.

For pH and specific gravity, summaries (1), (2) and (4) will be Analytical Method(s): provided.

> For each endpoint other than pH and specific gravity, summaries (3) and (4) will be provided.

(1) Summary of Urine Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided by subject type for each visit.

(2) Case Plots

Plots over time for each subject will be presented.

Number of Subjects in Categories of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided by subject type.

Property of Takedai. For not (4) Summary of Shifts of Urine Laboratory Test Results Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided by subject type.

For each urine laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

#### 6.8.3 Vital Signs, Weight and Height

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): Systolic Blood Pressure Diastolic Blood Pressure

> Heart Rate **Body Temperature**

Weight Height

**BMI** Respiration Rate

Visit: Using the (Baseline to Week 22) of the visit window defined in

Section 9.2.2.

For each endpoint, summaries (1) and (2) will be provided. Analytical Method(s):

(1) Summary of Vital Signs, Weight and Height, and Change from

Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - Baseline) will be provided by

subject type for each visit.

(2) Case Plots

Plots over time for each subject will be presented.

#### 6.8.4 **ECGs**

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): Heart Rate

PR Interval
PR Interval
QRS Interval
QT Interval
QTcF II-

[Within Normal Limits, Abnormal but not

Clinically Significant, Abnormal and

Clinically Significant]

Using the (Baseline to Week 22) of the visit window defined in

Analytical Method(s): For each endpoint other than 12-lead ECG interpretations, summaries

(1) and (2) will be provided.

For ECG interpretation, summary (3) will be provided.

- (1) Summary of ECG Parameters and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline (each post-baseline visit Baseline) will be provided by subject type for each visit.
- (2) Case Plots
  Plots over time for each subject will be presented
- (3) Summary of Shift of ECG Interpretation
  Shift table showing the number of subjects in each category at baseline and each post-baseline visit will be provided by subject type.

### 6.8.5 Displays of Treatment-Emergent Adverse Events (Japanese)

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): TEAE

Analytical Method(s): TEAEs will be summarized in the same way as in Section 6.8.1.2. All

summaries will be presented in Japanese.

### 6.9 Pharmacokinetic, Pharmacodynamic, and Biomarker Analyses

### 6.9.1 Pharmacokinetic Analysis

#### 6.9.1.1 Plasma Concentrations

Analysis Set: Safety Analysis Set

Analysis Endpoint(s): Plasma concentrations of TAK-625

Visit: Using the visits of the visit window defined in Section 9.2.2.

Analytical Method(s): The following summaries will be provided.

(1) Summary of Plasma Concentrations by Visit

Descriptive statistics will be provided by subject type by visit by
dose level categories administered just before sample collection.

\*\*A SAS Program for the WHO Growth \*\*Line \*\*A SAS Program for the WHO Growth \*\*Line \*\*India \*\*A SAS Program for the 2000 CDG \*\*Constant \*\*Const

JDI applicable applicable

There was no change to the protocol planned analyses.

#### 9.0 **APPENDIX**

#### 9.1 **Changes From the Previous Version of the SAP**

From the SAP version 1.0, the major updates except minor updates like error correction were following parts. ial use only and following parts.

Section 6.0 STATISTICAL ANALYSIS

Before the change

Not applicable.

After the change

Statistical analyses will be performed using all subjects' data up to Week 22 (i.e., up to Day 169 or 25OCT2023) after the data are locked. PK analysis will be performed using all subjects' data up to Week 12 after the data are locked.

Reason for the change

To make the target range of the Interim analysis clear.

Section 6.1 General Considerations

Before the change

- Descriptive statistics: Number of subjects, mean, standard deviation, standard error, maximum, minimum, and quartiles (Q1, median, and Q3).
- Duration of exposure to study drug (days): Date of last dose of study drug date of first dose of study drug + 1.
- Duration of study after baseline (days): Date of last visit/contact date of first dose of study drug + 1.

Kerms of Use Time to liver-associated events: PEBD surgery, listing for liver transplantation, liver decompensation [hepatic encephalopathy, variceal bleeding, ascites, and spontaneous bacterial peritonitis] events, hepatocellular carcinoma (HCC), death.

#### After the change

- Descriptive statistics for endpoints other than PK: Number of subjects, mean, standard deviation, standard error, maximum, minimum, and quartiles (Q1, median, and Q3).
- Descriptive statistics for PK: Number of subjects, mean, standard deviation, maximum, median, and minimum.
- Duration of exposure to study drug (days): {Date of last dose of study drug or Week 22 visit (ie. the latest visit by Day 169) which comes faster - date of first dose of study drug} + 1.
- Duration of study after baseline (days): {Date of last visit/contact or Week 22 visit (ie, the latest visit by Day 169) which comes faster - date of first dose of study drug} + 1.

Dose Level (μg/kg): Strength of study drug taken (mg) / (last available body weight (kg) prior to or on the day of study drug taken) \* 1000.

Dose Level Categories for PK (µg/kg): Categorize by following below calculation rule. If Min  $\leq$  dose level  $\leq$  300 µg/kg, then dose level category = 200 µg/kg; if 300 µg/kg  $\leq$  dose level  $\leq$  Max, then dose level category = 400  $\mu$ g/kg.

- Total Drug Exposure (µg/kg): Sum of {number of study drugs taken \* dose level received  $(\mu g/kg)$ .
- Average Daily Dose (µg/kg/day): Total Drug Exposure (µg/kg) / Duration of exposure to study drug (days).

Time to liver-associated events: PEBD surgery, listing for liver transplantation, liver decompensation [hepatic encephalopathy, variceal bleeding, ascites, and spontaneous bacterial peritonitis] events, hepatocellular carcinoma (HCC), death, and other.

Corrected Sodium (mEq/L): sodium (mEq/L) + (0.002 \* Triglycerides (mg/dL)).

- giagnosis of ALGS + 1) / 30.44.

  Significant Protocol Deviation: Deviation defined in the PDMP as "Important PD" whose Severity Classifications is "major" or "critical".

  Ison for the change ne calculation rules and definitions were added and updated.

  tion 6.1 General Considerations ore the change applicable.

  It the change ne reporting derived values or parameters. fall and the position of the

Reason for the change

Some calculation rules and definitions were added and updated.

Section 6.1 General Considerations

Before the change

Not applicable.

After the change

When reporting derived values or parameters, following presenting rules will be applied.

- For sBA, ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.
  - For measures of median and mean, use 3 decimal places.
  - For measures of standard deviation, standard error of the mean and CI, use 4 decimal places.
  - For measures of minimum and maximum values as well as observed value (for Listing), use 2 decimal places.
  - >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
  - For p-values use 3 decimal places.
  - Presentation of p-values display p-values that would round to 0.000 as <0.001.
- Other than sBA, and ItchRO: For rules on rounding and decimal presentation of these statistics, along with the rules for presenting certain derived values see below.
  - For measures of median and mean, use 1 decimal place beyond those used for the measurement.
  - For measures of standard deviation, standard error of the mean and CI, use 2 decimal places beyond those used for the measurement.
  - For measures of minimum and maximum values, use the same number of decimal places as those used for the measurement.
  - >=5 is rounded up away from zero, whereas <5 is rounded down toward zero, to account for rounding of negative numbers.
  - For p-values use 3 decimal places.

- Presentation of p-values display p-values that would round to 0.000 as <0.001.
- BMI should be rounded to 1 decimal place for reporting.
- Derived questionnaire scores, and other similar efficacy parameters recorded as integers should be rounded to 1 decimal place for reporting.
- Averaged lab results (e.g. Diastolic/Systolic Blood Pressure and Pulse [when taken in the applicable triplicate]) should be rounded to 1 decimal place for reporting.

Reason for the change

Presenting rules in TLF were added.

Section 6.2.1 Analysis Approach for Continuous Efficacy Endpoints

Before the change

- Change from Week 18 to Week 22:
  - ♦ Descriptive statistics and two-sided 95% confidence interval of mean will be provided for observed values (Week 18 and Week 22) and changes from Week 18 (Week 22 -Week 18). For endpoint with multiple visits, these will be provided by visit.
- Change from baseline to post-baseline:

Descriptive statistics and two-sided 95% confidence interval of mean will be provided for observed values (baseline and post-baseline visits) and changes from baseline (each postbaseline visit - baseline). For endpoint with multiple visits, these will be provided by visit.

After the change

- Change from Week 18 to Week 22:
  - ♦ Descriptive statistics and two-sided 95% confidence interval of mean will be provided for observed values (Week 18 (LOCF) and Week 22) and changes from Week 18 (Week 22 - Week 18 (LOCF)) by subject type. For endpoint with multiple visits, these will be provided by visit.
- Change from baseline to post-baseline:

Descriptive statistics and two-sided 95% confidence interval of mean will be provided for observed values (baseline and post-baseline visits) and changes from baseline (each postbaseline visit - baseline) by subject type. For endpoint with multiple visits, these will be provided by visit.

Reason for the change

To make it clear that LOCF visit will be used. For subject type, 2 analysis (without subject less than 1 year or with the one) will be planed as subject less than 1 year old was enrolled. Same change will be omitted hereafter.

Section 6.3.2 Screen Failures

Before the change

Analysis Endpoint(s): Age (months)

After the change

Not applicable.

Reason for the change

No infant subjects who failed screening.

Section 6.3.5 Disposition of Subjects

Before the change

w the applicable Terms of Use Analysis Endpoint(s): Study Drug Administration Status, [Eligible but Not Treated]

Reason for Not Being Treated, [AE, Screen Failure (Did not meet inclusion criteria or did meet exclusion criteria), Protocol Deviation, Lost to Follow-up, Pregnancy, Withdrawal by Subject, Study Terminated by Sponsor, Other]

Study Drug Completion Status, [Completed Study Drug, Prematurely Discontinued Study Drug]

Completion Status of All Planned Study Visits, Completed Study, Prematurely Discontinued Study]

Analytical Method(s): Frequency distributions will be provided. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the study drug will be used as the denominator. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

After the change

Analysis Endpoint(s):

Study Drug Completion Status, [Ongoing, Completed Study Drug, Prematurely Discontinued Study Drug

Completion Status of All Planned Study Visits, [Ongoing, Completed Study, Prematurely Discontinued Study]

Analytical Method(s): Frequency distributions will be provided by subject type. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

Reason for the change

Deleted analysis endpoints were not appropriate for ITT population. The category of "Ongoing" was added because this SAP is for Interim analysis.

### Section 6.3.6.1 Significant Protocol Deviations

Before the change

Analysis Endpoint(s): Significant Protocol Deviations, [AE, Screen Failure (Did not meet inclusion criteria or did meet exclusion criteria), Protocol Deviation, Lost to Follow-up, Pregnancy, Withdrawal by Subject, Study Terminated by Sponsor, Other]

After the change

Analysis Endpoint(s): Significant Protocol Deviations, [Informed Consent and Process, Inclusion Criteria, Exclusion Criteria, Concomitant Medication, Laboratory Assessment, Study Procedures (not safety and efficacy related), Safety, Visit Schedule, IP conditions, IP preparation, IP administration, Subject IP Compliance, Efficacy, Subject Discontinuation, Administrative, Patient Reported Outcomes, PK/PD, Other Criteria]

Reason for the change

Change it from CRF category to CTMS category.

Section 6.4.1 Demographic and Baseline Characteristics

Before the change

. . .

Analysis Endpoint(s): ItchRO(Obs) <u>4-week</u> Morning Average Severity (Item 1) Score, ItchRO(Obs) <u>4-week</u> Morning Average Frequency (Item 3) Score

After the change

. . .

Analysis Endpoint(s): ItchRO(Obs) <u>Weekly</u> Morning Average Severity (Item 1) Score, ItchRO(Obs) <u>Weekly</u> Morning Average Frequency (Item 3) Score

Reason for the change

Added CTD analysis category. Error correction.

Section 6.6 Extent of Exposure and Compliance

Before the change

Analysis Endpoint(s): Not applicable.

Analytical Method(s): (1) Study Drug Exposure and Compliance

Frequency distributions for categorical endpoints and descriptive statistics for continuous endpoints will be provided.

After the change

Analysis Endpoint(s): Total Drug Exposure (µg/kg), Average Daily Dose (µg/kg/day)

Analytical Method(s): (1) Study Drug Exposure, Compliance, <u>Total Drug Exposure and Average Daily Dose</u>

Frequency distributions for categorical endpoints and descriptive statistics for continuous endpoints will be provided by subject type.

Reason for the change

Added additional endpoints.

Section 6.7.4 Subgroup Analysis

Before the change

Subgroup(s): Age, [Min<= - <2, 2<= - <=4, 5<= - <=8, 9<= - <=12, 13<= - <=18, 18<- <=Max]

After the change

Subgroup(s): Age, [Min $\leq$  -  $\leq$  - < -

Reason for the change

To be consistent with CTD analysis.

Section 6.9.1.1 Plasma Concentrations

Before the change

Analytical Method(s): The following summaries will be provided.

(1) Summary of Plasma Concentrations by Visit Descriptive statistics will be provided.

After the change

Analytical Method(s): The following summaries will be provided.

(1) Summary of Plasma Concentrations by Visit Descriptive statistics will be provided by subject type by visit by dose level categories administered just before sample collection.

Reason for the change

To incorporate new Clinical pharmacology insight.

#### Section 9.2.1 Definition of Study Days

Before the change

The following definitions and calculation formulas will be used.

- Study Day: The day before the first dose of the study drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. If the date of the observation is on the same date or after the day of the first dose, Study Day will be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.
- Follow-up Day: The day after the last dose of the study drug will be defined as Follow-up Day 1. Follow-up Day will be calculated relative to Day 1.

After the change

The following definitions and calculation formulas will be used.

- Study Day: The day before the first dose of the study drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. If the date of the observation is on the same date or after the day of the first dose, Study Day will be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.
- Follow-up Day: The day after the last dose of the study drug will be defined as Follow-up Day 1.

Reason for the change

Error correction.

### Section 9.2.2.1 Endpoints other than ItchRO Scores and PK Samples

Before the change

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used.

After the change

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used. For laboratory test data, if there are two observations of both central laboratory sample and local sample on the same date, central laboratory sample data will be used. Values less than or equal to the lower limit of quantification

applicable Terms of Use will be treated as one-half of the lower limit value when calculating the descriptive statistics. Values greater than or equal to the upper limit of quantification will be treated as the upper limit value when calculating the descriptive statistics.

Reason for the change

Added handling rule for the lower limit of quantification value.

#### Section 9.2.2.2 PK Samples

Before the change

Study Time (hour) is defined as the difference from the PK sampling time at the visit date to the time of study drug taken at the visit date (rounded to 1 decimal place(s)).

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Time to the scheduled Study Time will be used. If there are two observations equidistant to the scheduled Study Time, the earlier observation will be used.

Table 9.9 Visit Window of PK

| Visit | D | ed Study<br>ay | Time Interval (days) Study Day | Scheduled Study<br>Time | Study<br>Time<br>(hours) |
|---|---|---|---|---|---|
| Pre-dose at Week 12 | Study<br>Day | 8.5 | <u>85</u> | Study 0<br>Time<br>(hour): | -5.0 ~<br>0.0 |
| 4 Hours after<br>Morning Dose at<br>Week 12 | Study<br>Day: | | <u>85</u> | Study 4<br>Time<br>(hour): | 3.0 ~ 5.0 |

After the change

Study Time (hour) is defined as the difference from the PK sampling time at the visit date to the time of study drug taken at the visit date (rounded to 1 decimal place(s)).

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Time to the scheduled Study Time will be used. If there are two observations equidistant to the scheduled Study Time, the earlier observation will be used. Values less than the lower limit of quantification will be treated as zero when calculating the descriptive statistics.

| Visit | D | ed Study<br>ay<br>ys) | Time Interval<br>(days)<br>Study Day | Scheduled Study<br>Time | Study<br>Time<br>(hours) |
|---|---|---|---|---|---|
| Pre-dose at Week 12 | Study<br>Day: | | <u>64 – 106</u> | Study 0 Time (hour): | -5:0 ~<br>0.0 |
| 4 Hours after<br>Morning Dose at<br>Week 12 | Study<br>Day: | | <u>64 – 106</u> | Study 4 Time (hour) | 3.0 ~ 5.0 |

Reason for the change

Added handling rule for the lower limit of quantification value. For Visit window, Time interval was update because previous interval was too narrow and inappropriate.

### Section 9.2.2.3 ItchRO Weekly Average Scores

#### Before the change

For visits other than LOCF visits [Week 18 (LOCF) and Week 48 (LOCF)], weekly average scores are calculated as the average of the scores (morning, evening, daily average of morning and evening, or daily maximum of morning and evening) over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). For the change from baseline calculations in weekly average ItchRO scores, baseline is defined in Table 9.10. Post-baseline weekly average ItchRO scores are only computed if at least 4 of the 7 daily ItchRO scores for the 7-day period are available. The restriction is not set for baseline ItchRO average scores.

In the event that a subject/caregiver failed to complete the morning/evening report, the morning/evening score for that day will be treated as missing data.

For each LOCF visit [Week 18 (LOCF) and Week 48 (LOCF)], if a subject/caregiver is not compliant with reporting ItchRO assessments during the 7-day period on or before the visit, the weekly average score from the most recent, previous compliant 7-day period will be used in a LOCF format. This process will be repeated as necessary. For example, if the 7-day period on or before the Week 18 (LOCF) visit (e.g., Study Days 120-126) is non-compliant, then Study Days 113-119 would be used.

#### After the change

For visits other than LOCF visits [Week 18 (LOCF)], weekly average scores are calculated as the average of the scores (morning, evening, daily average of morning and evening, or daily

maximum of morning and evening) over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). For the change from baseline calculations in weekly average ItchRO scores, baseline is defined in Table 9.10. Post-baseline weekly average ItchRO scores are only computed if at least 4 of the 7 daily ItchRO scores for the 7-day period are available. The restriction is not set for baseline ItchRO average scores.

In the event that a subject/caregiver failed to complete the morning/evening report, the morning/evening score for that day will be treated as missing data.

For each LOCF visit [Week 18 (LOCF)], if a subject/caregiver is not compliant with reporting ItchRO assessments during the 7-day period on or before the visit, the weekly average score from the most recent, previous compliant 7-day period will be used in a LOCF format. This process will be repeated as necessary. For example, if the 7-day period on or before the Week 18 (LOCF) visit (e.g., Study Days 120-126) is non-compliant, then Study Days 113-119 would be

Section 9.2.2.4 ItchRO 4-week Average Scores of Warld Subjection 9.2.2.4 ItchRO 4-week Average Scores of Warld Subject of Scores are calculated and even of the scores are calculated and even of the scores are calculated and even of the scores are calculated and even of the scores are calculated and even of the scores are calculated as a score of the scores are calculated as a score of the scores are calculated as a score of the scores are calculated as a score of the scores are calculated as a score of the For visits other than LOCF visits [Week 18 (LOCF) and Week 48 (LOCF)], 4-week average scores are calculated as the average of the scores (morning, evening, daily average of morning and evening, or daily maximum of morning and evening) over the visit consisting of the 28 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of nonmissing scores). For the change from baseline calculation in 4-week average ItchRO scores, baseline is defined in Table 9.11. Post-baseline 4-week average ItchRO scores are only computed if at least 20 of the 28 daily ItchRO scores for the 28-day period are available. The restriction is not set for baseline ItchRO average scores.

In the event that a subject/caregiver failed to complete the morning/evening report, the morning/evening score for that day will be treated as missing data.

For each LOCF visit [Week 18 (LOCF) and Week 48 (LOCF)], if a subject/caregiver is not compliant with reporting ItchRO assessments during the 28-day period on or before the visit, the 4-weekly average score from the most recent, previous compliant 28-day period will be used in a LOCF format, where the 28 days minus the 7 days immediately prior to the study visit will be used. This process will be repeated as necessary. For example, if the 28-day period on or before the Week 18 (LOCF) visit (e.g., Study Days 99-126) is non-compliant, then Study Days 92-119 would be used.

After the change

For visits other than LOCF visits [Week 18 (LOCF)], 4-week average scores are calculated as the average of the scores (morning, evening, daily average of morning and evening, or daily maximum of morning and evening) over the visit consisting of the 28 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). For the change from baseline calculation in 4-week average ItchRO scores, baseline is defined in Table 9.11. Post-baseline 4-week average ItchRO scores are only computed if at least 20 of the 28 daily ItchRO scores for the 28-day period are available. The restriction is not set for baseline ItchRO average scores.

In the event that a subject/caregiver failed to complete the morning/evening report, the morning/evening score for that day will be treated as missing data.

For each LOCF visit [Week 18 (LOCF)], if a subject/caregiver is not compliant with reporting ItchRO assessments during the 28-day period on or before the visit, the 4-weekly average score from the most recent, previous compliant 28-day period will be used in a LOCF format, where the 28 days minus the 7 days immediately prior to the study visit will be used. This process will be repeated as necessary. For example, if the 28-day period on or before the Week 18 (LOCF) visit (e.g., Study Days 99-126) is non-compliant, then Study Days 92-119 would be used. use only and

Reason for the change

Error correction.

Section 9.2.3 Partial Date Conventions

Before the change

Not applicable.

After the change

### 9.2.3 Partial Date Conventions

For Medication History and Concomitant Medication, if their stop date is partially/completely missing, following handling rules will be applied.

if (CMCAT="MEDICATION HISTORY") then "(1) Prior Medication";

else if (CMENRTPT="ONGOING") then "(3) Concomitant Medication";

else if

```
medication end year < TAK-625 start year) or
  medication end year = TAK-625 start year and
< medication end month < TAK-625 start month) or
  medication end year = TAK-625 start year and
  medication end month = TAK-625 start month and
```

< medication end date < TAK-625 start date ) then "(2) Concomitant Medication";

### else "(3) Concomitant Medication";

Reason for the change

To make it clear how to handle partial date.

#### 9.2 **Data Handling Conventions**

#### 9.2.1 **Definition of Study Days**

The following definitions and calculation formulas will be used.

- the applicable Terms of Use offine Study Day: The day before the first dose of the study drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. If the date of the observation is on the same date or after the day of the first dose, Study Daywill be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.
- Follow-up Day: The day after the last dose of the study drug will be defined as Follow-up Day 1.

# Definition of Study Visit Windows 9.2.2

When calculating Study Day relative to a reference date (ie, date of first dose of study drug [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0.

When calculating Follow-up Day relative to a reference date (ie. date of last dose of study drug [Follow-up Day 0]), it will be calculated as: date of observation - reference date. Hence, reference day is always Follow-up Day 0.

All evaluable data (ie, non-missing data) will be handled according to the following rules.

#### 9.2.2.1 Endpoints other than ItchRO Scores and PK Samples

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used. For laboratory test data, if there are two observations of both central laboratory sample and local sample on the same date, central laboratory sample data will be used. Values less than or equal to the lower limit of quantification will be treated as one-half of the lower limit value when calculating the descriptive statistics. Values greater than or equal to the upper limit of quantification will be treated as the upper limit value when calculating the descriptive statistics.

Table 9.1 Visit Window of sBA

| | Scheduled Study Day<br>(days) | | Time Interval (days) | |
|---|---|---|---|---|
| Visit | | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: | 1 | -42 - 1 | 10) |
| Week 12 | Study Day: | 85 | 2 - 106 | <15 |
| Week 18 | Study Day: | 127 | 107 - 141 | <b>≥</b> 15 |
| Week 22 | Study Day: | 155 | 142 - 169 | <15 |
| Week 18 (LOCF) | Study Day: | 127 | 2 - 141 | <15 |

Table 9.2 Visit Window of Liver Enzymes (ALT, ALP) and Bilirubins (Total and Direct)

| | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -42 - 1 | |
| Week 3 | Study Day: 22 | 2 - 32 | <15 |
| Week 6 | Study Day: 43 | 33 - 64 | <15 |
| Week 12 | Study Day: 85 | 65 - 106 | <15 |
| Week 18 | Study Day: 127 | 107 - 141 | <15 |
| Week 22 | Study Day: 155 | 142 - 169 | <15 |
| Week 18 (LOCF) | Study Day: 127 | 2 - 141 | <15 |

Table 9.3 Visit Window of Vital Signs, Weight and Height,

CBC, Coagulation, Chemistry Panel,
Urinalysis, Serum Storage Samples

| . 10 | Scheduled Study Day | | Time Interval (days) | |
|---|---|---|---|---|
| Visit | (days) | | | Follow-up Day |
| Baseline (Week 0) | Study Day: | 1 | -42 - 1 | |
| Week 3 | Study Day: | 22 | 2 - 32 | <15 |
| Week 6 | Study Day: | 43 | 33 - 64 | <15 |
| Week 12 | Study Day: | 85 | 65 - 106 | <15 |
| Week 18 | Study Day: | 127 | 107 - 141 | <15 |
| Week 22 | Study Day: | 155 | 142 - 169 | <15 |



Table 9.5 Visit Window of ECGs

| | Scheduled Study Day | | Time Inter | val (days) |
|-------------------|---------------------|----|------------|---------------|
| Visit | (days) | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: | 1 | -42~1 | |
| Week 12 | Study Day: | 85 | Q - 141 | <15 |



Table 9:8 Visit Window of Lipid Panel, Cholestasis Biomarkers (sBA subspecies, C4, FGF19), Lipid Soluble Vitamins

| O | Scheduled Study Day | | Time Interval (days) | |
|---|---|---|---|---|
| Visit | (days) | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: | 1 | -42 - 1 | |
| Week 12 | Study Day: | 85 | 2 - 106 | <15 |
| Week 18 | Study Day: | 127 | 107 - 141 | <15 |
| Week 22 | Study Day: | 155 | 142 - 169 | <15 |

#### 9.2.2.2 PK Samples

Study Time (hour) is defined as the difference from the PK sampling time at the visit date to the time of study drug taken at the visit date (rounded to 1 decimal place(s)).

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Time to the scheduled Study Time will be used. If there are two observations equidistant to the scheduled Study Time, the earlier observation will be used. Values less than the lower limit of quantification will be treated as zero when calculating the descriptive statistics.

| 1 able 9.9 | VISIT WINDOW OF PK |
|------------|--------------------|

| Visit | Scheduled Stu<br>(days) | dy Day | Time Interval<br>(days)<br>Study Day | Scheduled St | udy Time | Study<br>Time<br>(hours) |
|---|---|---|---|---|---|---|
| Pre-dose at Week 12 | Study Day: | 85 | 64 - 106 | Study Time<br>(hour): | 0 | <b>-5.0</b> ∼ <b>0.0</b> |
| 4 Hours after Morning<br>Dose at Week 12 | Study Day: | 85 | 64 - 106 | Study Time<br>(hour): | 4 | 3.0 ~ 5.0 |

## 9.2.2.3 ItchRO Weekly Average Scores

For visits other than LOCF visits [Week 18 (LOCF)], weekly average scores are calculated as the average of the scores (morning, evening, daily average of morning and evening, or daily maximum of morning and evening) over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). For the change from baseline calculations in weekly average ItchRO scores, baseline is defined in Table 9.10. Post-baseline weekly average ItchRO scores are only computed if at least 4 of the 7 daily ItchRO scores for the 7-day period are available. The restriction is not set for baseline ItchRO average scores.

In the event that a subject/caregiver failed to complete the morning/evening report, the morning/evening score for that day will be treated as missing data.

For each LOCF visit [Week 18 (LOCF)], if a subject/caregiver is not compliant with reporting ItchRO assessments during the 7-day period on or before the visit, the weekly average score from the most recent, previous compliant 7-day period will be used in a LOCF format. This process will be repeated as necessary. For example, if the 7-day period on or before the Week 18 (LOCF) visit (e.g., Study Days 120-126) is non-compliant, then Study Days 113-119 would be used.

| | Scheduled Study Day<br>(days) | | Time Inter | val (days) |
|---|---|---|---|---|
| Visit | | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: | -1 | -71 | 10/1 |
| Week 3 | Study Day: | 21 | 15 - 21 | <15 |
| Week 6 | Study Day: | 42 | 36 - 42 | O-15 |
| Week 12 | Study Day: | 84 | 78 - 84 | <15 |
| Week 18 | Study Day: | 126 | 120 - 126 | <15 |
| Week 19 | Study Day: | 133 | 127 - 133 | <15 |
| Week 20 | Study Day: | 140 | 134 - 140 | <15 |
| Week 21 | Study Day: | 147 | 141 - 147 | <15 |
| Week 22 | Study Day: | 154 | • 148 - 154 | <15 |
| Week 18 (for LOCF and<br>Responder Analysis) | Study Day: | 126 | 1 - 126 | <15 |

Table 9.10 Visit Window of ItchRO Weekly Average Score

### 9.2.2.4 ItchRO 4-week Average Scores

For visits other than LOCF visits [Week 18 (LOCF)], 4-week average scores are calculated as the average of the scores (morning, evening) daily average of morning and evening, or daily maximum of morning and evening) over the visit consisting of the 28 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). For the change from baseline calculation in 4-week average ItchRO scores, baseline is defined in Table 9.11. Post-baseline 4-week average ItchRO scores are only computed if at least 20 of the 28 daily ItchRO scores for the 28-day period are available. The restriction is not set for baseline ItchRO average scores.

In the event that a subject/caregiver failed to complete the morning/evening report, the morning/evening score for that day will be treated as missing data.

For each LOCE visit [Week 18 (LOCF)], if a subject/caregiver is not compliant with reporting ItchRO assessments during the 28-day period on or before the visit, the 4-weekly average score from the most recent, previous compliant 28-day period will be used in a LOCF format, where the 28 days minus the 7 days immediately prior to the study visit will be used. This process will be repeated as necessary. For example, if the 28-day period on or before the Week 18 (LOCF) visit (e.g., Study Days 99-126) is non-compliant, then Study Days 92-119 would be used.

| | Scheduled Study Day | | Time Int | erval (days) |
|-------------------|---------------------|-----|-----------|---------------|
| Visit | (days) | | | Follow-up Day |
| Baseline (Week 0) | Study Day: | -1 | -281 | 10 |
| Week 6 | Study Day: | 42 | 15 - 42 | <15 |
| Week 12 | Study Day: | 84 | 57 - 84 | <b>1</b> 5 |
| Week 18 | Study Day: | 126 | 99 - 126 | × <0 <15 |
| Week 22 | Study Day: | 154 | 127 - 154 | <15 |
| Week 18 (LOCF) | Study Day: | 126 | 1 - 126 | <b>⊘</b> <15 |

Table 9.11 Visit Window of ItchRO 4-week Average Score

#### 9.2.3 Partial Date Conventions

For Medication History and Concomitant Medication, if their stop date is partially/completely missing, following handling rules will be applied.

#### 9.3 Derivation of Endpoints

## 9.3.1 Change from Week 18 to Week 22 of Primary and Secondary Efficacy Endpoints

For each endpoint (primary and secondary efficacy endpoints), the change from Week 18 to Week 22 of the endpoint is defined as the difference between a value at Week 22 and a value at Week 18 (LOCF).

#### 9.3.2 ItchRO Average Scores

Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe (Item 1) or more frequent (Item 3) itching.

- ItchRO(Obs/Pt) Weekly Average Morning Score: Sum of ItchRO daily morning scores (over a 7-day period) divided by the number of days ItchRO completed. The definition applies to both severity (Item 1) weekly average scores.
- ItchRO(Obs/Pt) Weekly Average Severity Score (based on the daily maximum of morning and evening scores): Sum of ItchRO(Obs) daily maximum of morning and evening scores (over a 7-day period) divided by the number of days ItchRO completed.
- ItchRO (Obs/Pt) Weekly Average Severity Score (based on the daily average of morning and evening scores): Sum of ItchRO(Obs) daily average of morning and evening scores (over a 7-day period) divided by the number of days ItchRO completed.
- ItchRO(Obs/Pt) 4-Week Average Morning Score: Sum of ItchRO daily morning scores (over a 28-day period) divided by the number of days ItchRO completed. The definition applies to both severity (Item 1) and frequency (Item 3, Observer only) 4-week average scores.
- ItchRO(Obs/Pt) 4-Week Average Evening Score: Sum of ItchRO daily evening scores (over a 28-day period) divided by the number of days ItchRO completed. The definition applies to both severity (Item 1) and frequency (Item 3, Observer only) 4-week average scores.





Z-scores of weight, height and BMI are based on a subject's gender and age at each scheduled visit. For subjects less than 24 months of age, the World Health Organization (WIII) and the charts are recommended by the Commended b charts are recommended by the Centers for Disease Control (CDC) and will be used to derive z-scores. For subjects at least 24 months of age, the CDC growth charts will be used to derive z-scores.

ror calculated to the state of Age at which height and weight were measured should be used for calculating z-scores, not using

### 9.3.6 Lists of Laboratory Tests

| H(CDC '41 | Charita | T * .* 1 D 1 | TI da a banda |
|---|---|---|---|
| Hematology (CBC with Differential) | <u>Chemistry</u> | <u>Lipid Panel</u> | <u>Urinalysis</u> |
| · | Albumin | Total cholesterol | pH |
| Hematocrit | ALP | LDL-C (direct) | Specific gravity Protein Glucose |
| Hemoglobin | Amylase | HDL-C | Protein |
| MCV, MCH, MCHC | ALT (SGPT) | TG | Glucose |
| Red blood cells | AST (SGOT) | | Ketones |
| Platelets | Bicarbonate | Cholestasis Biomarkers <sup>a</sup> | Bilirubin |
| White blood cells | Bilirubin, direct | sBA (LC-MS) | Occult blood and cells |
| WBC Differential (% and | (conjugated) | sBA subspecies | Nitrite |
| absolute) | Total serum Bilirubin | 7alpha-C4 | Urobilinogen |
| Neutrophils | (TSB) | FGF-19 | Leukocyte esterase |
| Eosinophils | BUN | Autotaxin | Microscopic examination |
| Basophils | Calcium | 200 | Oxalate |
| Lymphocytes | Chloride | Lipid Soluble | Urinary creatinine |
| Monocytes | Creatinine | Vitamins S | ormary creatinine |
| | GGT | 25-hydroxy vitamin D | |
| <b>Coagulation</b> | Glucose | Retinol | |
| aPTT (sec) | Lipase | RBP | |
| INR | Phosphate | Alpha-tocopherol | |
| PT (sec) | Potassium | Estimated Total Lipids | |
| | Sodium | Ratio of Alpha-tocopherol | |
| | Corrected Sodium | to Estimated Total Lipids | |
| | Total protein | - | |
| | Total sBA (enzymatic assay) | | |
| | Uric Acid | | |
| | Measured serum<br>Osmolality | | |

# 9.3.7 Table for AECI

The categories of AECI will follow ones in CRF.

# 9.3.8 Significance Level and Confidence Coefficient

Significance level: 5% (two-sided).

• Confidence coefficient: 95% (two-sided).

## 9.4 Analysis Software

SAS (version 9.4)